CLINICAL TRIAL: NCT04435626
Title: A Multicenter, Randomized, Double-blind, Parallel-group, Placebo-controlled Study to Evaluate the Efficacy and Safety of Finerenone on Morbidity and Mortality in Participants With Heart Failure (NYHA II-IV) and Left Ventricular Ejection Fraction ≥ 40% (LVEF ≥ 40%)
Brief Title: Study to Evaluate the Efficacy (Effect on Disease) and Safety of Finerenone in Participants With Heart Failure and Left Ventricular Ejection Fraction (Proportion of Blood Expelled Per Heart Stroke) Greater or Equal to 40%
Acronym: FINEARTS-HF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20103; 2020-000306-29 (EudraCT Number)
Record Dates: First submitted 2020-06-15; First posted 2020-06-17 (Actual); Results first posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure
Keywords: Heart Failure with Preserved Ejection Fraction,; Mineralocorticoid receptor antagonist (MRA)
MeSH Terms: conditions — Heart Failure | interventions — finerenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1_BAY94-8862 (Experimental): Adult patients receive BAY94-8862
  Interventions: Drug: Finerenone (BAY94-8862)
- Arm 2_Placebo (Placebo Comparator): Adult patients receive placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Finerenone (BAY94-8862) — For participants with an eGFR ≤60 mL/min/1.73 m^2: Starting dose is 10 mg OD and maximum dose 20 mg OD.
  For participants with an eGFR >60 mL/min/1.73 m^2: Starting dose is 20 mg OD and maximum dose 40 mg OD. Finerenone is administered orally as immediate release tablets.
  Arms: Arm 1_BAY94-8862
Other: Placebo — Placebo tablets matching BAY94-8862 are administered orally.
  Arms: Arm 2_Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of finerenone compared to placebo (a tablet without active substance) in the reduction of cardiovascular death (generally meaning death due to disease of the heart or blood vessels) and total Heart Failure (HF) events, including HF hospitalization and urgent visits for HF(generally meaning a hospital stay or urgent presentation to a healthcare unit due to worsening symptoms of heart failure) in patients suffering from HF with an ejection fraction greater than or equal to 40%. Researchers will also collect information on how much the heart disease has impact on patient's lives, change of kidney function, and how well finerenone treatment is tolerated. The study plans to enroll 6000 male and female patients of the age of 40 years and above suffering from heart failure with ejection fraction greater than or equal to 40%. Participants will take the study product as oral tablet with a dose between 0 (Placebo) 40 mg once daily. Study duration will be up to 43 months.

ELIGIBILITY:
Inclusion Criteria:

* Participant (male or female) must be aged 40 years and older.
* Diagnosis of heart failure with New York Heart Association(NYHA) class II-IV, ambulatory or hospitalized primarily for heart failure.
* On diuretic treatment for at least 30 days prior to randomization.
* Documented left ventricular ejection fraction (LVEF) of ≥40% measured by any modality within the last 12 months.
* Structural heart abnormalities based on any local imaging measurement within the last 12 months, defined by at least one of the following findings: left atrial diameter (LAD) ≥3.8cm, left atrial area (LAA) ≥20cm2, left atrial volume index (LAVI) >30 mL/m2, left ventricular mass index (LVMI) ≥115 g/m2 (♂)/ 95 g/m2 (♀), septal thickness or posterior wall thickness ≥1.1 cm
* n-terminal prohormone B-type natriuretic peptide (NT-proBNP) ≥300 pg/mL (BNP ≥100 pg/mL) in sinus rhythm and patient does not have an ongoing diagnosis of paroxysmal atrial fibrillation or NT-proBNP ≥900 pg/mL (BNP ≥300 pg/mL) in atrial fibrillation (or if atrial fibrillation status is unknown or if patient has an ongoing diagnosis of paroxysmal atrial fibrillation) for participants obtained at the following time:

  * Within 90 days prior to randomization if patient had been hospitalized for heart failure (HF) requiring initiation or change in HF therapy or if patient had an urgent visit for HF requiring intravenous (IV) diuretic therapy, both within 90 days prior to randomization OR
  * Within 30 days prior to randomization if patient has not been hospitalized for HF nor had an urgent HF visit within the past 90 days.
* Women of childbearing potential can only be included in the study if a pregnancy test is negative at screening and baseline and if they agree to use adequate contraception which is consistent with local regulations regarding the methods for contraception for those participating in clinical trials.

Exclusion Criteria:

* Estimated glomerular filtration rate (eGFR) <25 mL/min/1.73 m² at either screening or randomization visit.
* Serum/plasma potassium >5.0 mmol/L at either screening or randomization visit.
* Acute inflammatory heart disease, e.g. acute myocarditis, within 90 days prior to randomization
* Myocardial infarction or any event which could have reduced the ejection fraction within 90 days prior to randomization
* Coronary artery bypass graft surgery in the 90 days prior to randomization
* Percutaneous coronary intervention in the 30 days prior to randomization
* Stroke or transient ischemic cerebral attack within 90 days prior to randomization
* Probable alternative cause of participants' HF symptoms that in the opinion of the investigator primarily accounts for patient's dyspnea such as significant pulmonary disease, anemia or obesity. Specifically, patients with the below are excluded: Severe pulmonary disease requiring home oxygen, or chronic oral steroid therapy, History of primary pulmonary arterial hypertension, Hemoglobin <10 g/dl, Valvular heart disease considered by the investigator to be clinically significant, Body Mass Index (BMI) >50 kg/m2 at screening
* Systolic blood pressure(SBP) ≥160 mmHg if not on treatment with ≥3 blood pressure lowering medications or ≥180 mmHg irrespective of treatments, on 2 consecutive measurements at least 2-minute apart, at screening or at randomization.
* Concomitant systemic therapy with potent cytochrome P450 isoenzyme 3A4 (CYP3A4) inhibitors (e.g. itraconazole, ritonavir, indinavir, cobicistat, clarithromycin) or moderate or potent CYP3A4 inducers, that cannot be discontinued 7 days prior to randomization and for the duration of the treatment period.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6016 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-06-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (661):
- United States (107):
  - Cardiology, PC, Birmingham, Alabama
  - Eastern Shore Research Institute, LLC | Fairhope, AL, Fairhope, Alabama
  - Mobile Heart Specialists - Providence, Mobile, Alabama
  - University of Arizona Clinical and Translational Sciences Research Center, Tucson, Arizona
  - Heart Clinic Arkansas, Little Rock, Arkansas
  - WestSide Medical, Beverly Hills, California
  - CA Heart and Vein Specialists, Huntington Beach, California
  - UCI Medical Center - Neurology, Orange, California
  - Sutter Medical Center - Cardiology, Sacramento, California
  - NorthBay Clinical Research, LLC | Santa Rosa, CA, Santa Rosa, California
  - The Lundquist Institute - Gynecology, Torrance, California
  - Blue Coast Research Center, LLC, Vista, California
  - Interventional Cardio Medical- DCT Department, West Hills, California
  - Interventional Cardiology Medical Group | West Hills, CA, West Hills, California
  - VA Eastern Colorado Health Care System, Aurora, Colorado
  - Colorado Springs Cardiology - Woodmen Medical Plaza, Colorado Springs, Colorado
  - South Denver Cardiology Associates, PC, Littleton, Colorado
  - Cardiovascular & Vein Center of Florida | Bradenton, FL, Bradenton, Florida
  - Nova Clinical Research - Blake Medical Center, Bradenton, Florida
  - Cardiology Associates Research Company, Daytona Beach, Florida
  - North Florida Foundation for Research and Education - Clinical Trial Center, Gainesville, Florida
  - LifeSpring Research Foundation, LLC, Miami, Florida
  - Southwest Florida Research | Naples, FL, Naples, Florida
  - East Coast Institute for Research | St. Augustine, FL, Saint Augustine, Florida
  - Cardiology Partners Clinical Research Institute | Wellington Office, Wellington, Florida
  - Centricity Research at Talbotton, Columbus, Georgia
  - Atlanta Heart Specialists - Tucker, Tucker, Georgia
  - Advocate Illinois Masonic Medical Center - Cardiology, Chicago, Illinois
  - Advocate Good Samaritan Hospital - Cardiology, Downers Grove, Illinois
  - Advocate Condell Medical Center, Libertyville, Illinois
  - Edward Hospital - Main Campus - Cardiology, Naperville, Illinois
  - Captain James A. Lovell Federal Health Care Center, North Chicago, Illinois
  - Carle Health Methodist Hospital - Cardiology, Peoria, Illinois
  - Midwest Cardiovascular Research and Education Foundation | Elkhart, IN, Elkhart, Indiana
  - Reid Physicians Associates - Cardiology Department, Richmond, Indiana
  - Kansas Nephrology Research Institute, Wichita, Kansas
  - Baptist Health Paducah - Cardiology, Paducah, Kentucky
  - Cardiovascular Associates Research, LLC, Covington, Louisiana
  - Heart Clinic of Hammond, Hammond, Louisiana
  - Louisiana Heart Center - Slidell, Slidell, Louisiana
  - Southern Clinical Research, LLC, Zachary, Louisiana
  - MaineHealth Cardiology - Scarborough, Scarborough, Maine
  - Johns Hopkins Hospital - Cardiology, Baltimore, Maryland
  - Suburban Hospital - Cardiology, Bethesda, Maryland
  - Cardiovascular Specialists of Central Maryland, PA, Columbia, Maryland
  - Henry Ford Hospital - OB/GYN, Detroit, Michigan
  - AA Medical Research Center | Flint, MI, Flint, Michigan
  - M Health Fairview Heart Clinic - Maplewood, Maplewood, Minnesota
  - M Health Fairview Heart Clinic - Fulton, Minneapolis, Minnesota
  - St. Cloud Hospital, Saint Cloud, Minnesota
  - Baptist Heart -Cardiology - DCT Dept, Jackson, Mississippi
  - University Hospital - UMMC - Nephrology, Jackson, Mississippi
  - Harry S Truman Memorial Veterans Hospital - Cardiology, Columbia, Missouri
  - Clinical Research Consultants, Kansas City, Missouri
  - Saint Luke's Mid America Heart Institute, Kansas City, Missouri
  - Mercy Hospital Springfield - Cardiology, Springfield, Missouri
  - Logan Health Research, Kalispell, Montana
  - CHI Health Clinic Heart Institute - Grand Island, Grand Island, Nebraska
  - CHI Health Nebraska Heart, Lincoln, Nebraska
  - Advanced Heart Care, LLC | Bridgewater, NJ, Bridgewater, New Jersey
  - NJ Heart | Linden, NJ, Linden, New Jersey
  - Garden State Heart Care, Manalapan, New Jersey
  - Nuvance Health - The Heart Center, Poughkeepsie, New York
  - Division of Cardiovascular Research at Peconic Bay Medical Center, Riverhead, New York
  - Laurelton Heart Specialists, Rosedale, New York
  - Saratoga Clinical Research, LLC, Saratoga Springs, New York
  - Cardiac Care & Vascular Medicine, The Bronx, New York
  - Northwell Health Physician Partners Cardiology at Valley Stream, Valley Stream, New York
  - Kernodle Clinic West, Burlington, North Carolina
  - University of North Carolina, Chapel Hill, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Kettering Health Network | Research Institute, Kettering, Ohio
  - Rama Research LLC | Marion, OH, Marion, Ohio
  - Mercy Health - St. Elizabeth Youngstown Hospital, Youngstown, Ohio
  - South Oklahoma Heart Research, LLC, Oklahoma City, Oklahoma
  - Capital Area Research | Camp Hill, PA, Camp Hill, Pennsylvania
  - Doylestown Health Cardiology - DCA, Doylestown, Pennsylvania
  - Kent Hospital, Warwick, Rhode Island
  - Trident Cardiology Associates, PA, Ladson, South Carolina
  - Carolina Heart Specialists | Lancaster, SC, Lancaster, South Carolina
  - Monument Health Clinical Research, Rapid City, South Dakota
  - Sanford USD Medical Center - Cardiology, Sioux Falls, South Dakota
  - The Stern Cardiovascular Foundation - Germantown, TN, Germantown, Tennessee
  - Apex Research Foundation, LLC. | Jackson, TN, Jackson, Tennessee
  - Lt. Col. Luke Weathers, Jr. VA Medical Center - Cardiology, Memphis, Tennessee
  - Cardiovascular Research of Knoxville, Powell, Tennessee
  - Ascension Seton Heart Specialty Care and Transplant Center, Austin, Texas
  - Texas Health & Vascular Specialists - Dallas, Dallas, Texas
  - Southwest Family Medicine Associates | Dallas, TX, Dallas, Texas
  - Texas Health Family Care - W Vickery Blvd, Fort Worth, Texas
  - University of Texas Medical Branch at Galveston, Galveston, Texas
  - Houston Heart & Vascular Associates, Humble, Texas
  - South Texas Cardiovascular Consultants, PLLC / Kerrville, TX, Kerrville, Texas
  - North Dallas Research Associates, McKinney, Texas
  - ClinRx Research, LLC, Plano, Texas
  - South Texas Cardiovascular Consultants - San Antonio, San Antonio, Texas
  - Clinical Advancement Center, PLLC, San Antonio, Texas
  - Northwest Houston Clinical Research - Tomball, Tomball, Texas
  - University of Utah Clinical Neurosciences Center, Salt Lake City, Utah
  - Inova Cardiology- Fairfax, Fairfax, Virginia
  - Virginia Heart, Falls Church, Virginia
  - Virginia Heart - Leesburg, Leesburg, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Salem VA Medical Center - Cardiology, Salem, Virginia
  - Selma Medical Associates, Winchester, Virginia
  - William S. Middleton Memorial Veterans Hospital, Madison, Wisconsin
  - Aurora Saint Luke's Medical Center - Cardiology, Milwaukee, Wisconsin
- Argentina (19):
  - Centro de Investigaciones Metabolicas | Ciudad de Autonoma de Buenos Aires, Argentina, Ciudad Autónoma de Buenos Aire, Buenos Aires
  - Clínica Coronel Suarez, Coronel Suárez, Buenos Aires
  - Hospital Italiano de La Plata | Clinical Research Department, La Plata, Buenos Aires
  - Centro de Investigaciones Medicas Lanus | Buenos Aires, Argentina, Lanús, Buenos Aires
  - Sanatorio Modelo Quilmes, Quilmes, Buenos Aires
  - Corporación Médica de General San Martín, San Martín, Buenos Aires
  - Instituto De Investigaciones Clinicas Zarate | Zarate, Argentina, Zárate, Buenos Aires
  - Instituto Cardiovascular de Buenos Aires | Buenos Aires, Argentina, Buenos Aires, Buenos Aires F.D.
  - Hospital Militar Central "CIR. MY. C. Argerich", Buenos Aires, Ciudad Auton. de Buenos Aires
  - Centro de Especialidades Medicas (CEMEDIC), Buenos Aires, Ciudad Auton. de Buenos Aires
  - CEDIC Centro de Investigación Clínica | Buenos Aires, Argentina, CABA, Ciudad Auton. de Buenos Aires
  - Grupo Orono | Instituto Cardiovascular de Rosario - Insuficiencia Cardiaca y Trasplante Department, Rosario, Santa Fe Province
  - Consultorios Integrados Rosario | Instituto Medico de la Fundacion de Estudios Clinicos, Rosario, Santa Fe Province
  - Instituto de Cardiologia | Tucuman, AR, San Miguel de Tucumán, Tucumán Province
  - Investigaciones Medicas IMOBA S.R.L., Buenos Aires
  - Instituto de Cardiologia de Corrientes Juana F. Cabral | Corrientes, Argentina, Corrientes
  - Clínica Privada del Prado, Córdoba
  - Instituto Médico DAMIC- Fundación Rusculleda, Córdoba
  - Centro de Investigaciones Clinicas del Litoral | Santa Fe, Argentina, Santa Fe
- Australia (10):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - The Wesley Hospital, Auchenflower, Queensland
  - The Prince Charles Hospital, Chermside, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Advara HeartCare Leabrook, Leabrook, South Australia
  - Advara HeartCare Ringwood, Bundoora, Victoria
- Austria (9):
  - Klinikum Klagenfurt am Wörthersee, Klagenfurt, Carinthia
  - Universitätsklinikum St. Pölten, Sankt Pölten, Lower Austria
  - Medizinische Universität Graz, Graz, Styria
  - Krankenhaus St. Josef Braunau | Innere Medizin I, Braunau am Inn, Upper Austria
  - Landeskrankenhaus Feldkirch, Feldkirch, Vorarlberg
  - Uniklinikum Salzburg - Landeskrankenhaus, Salzburg
  - Universitätsklinikum AKH Wien, Vienna
  - Imed19-privat, Vienna
  - Klinik Floridsdorf - Krankenhaus Nord, Vienna
- Brazil (19):
  - Santa Casa de Misericórdia da Bahia, Salvador, Estado de Bahia
  - Hospital do Coração do Brasil, Brasília, Federal District
  - Hospital das Clinicas da Universidade Federal de Goias | Centro de Pesquisa em Cardiologia, Goiânia, Goiás
  - Quanta Diagnostico Por Imagem | Research and Innovation Department, Curitiba, Paraná
  - Sociedade Hospitalar Angelina Caron | Departamento de Ensino e Pesquisa, Paraná, Paraná
  - Fundação Universidade de Caxias do Sul, Caxias do Sul, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre | Clinical Research Center - Surgery Research Center, Porto Alegre, Rio Grande do Sul
  - Hospital Mae de Deus, Porto Alegre, Rio Grande do Sul
  - FZ Pesquisa e Servicos em Cardiologia | Porto Alegre, Brazil, Porto Alegre, Rio Grande do Sul
  - MK Consultoria Médico Científica Ltda/Angiocor Blumenau, Blumenau, Santa Catarina
  - Centro de Pesquisa Clinica do Coração | Aracaju, Brasil, Aracaju, Sergipe
  - Hospital Felício Rocho, Belo Horizonte, São Paulo
  - Campinas Clinical Research Institute (IPECC) | Campinas, Brazil, Campinas, São Paulo
  - Instituto do Coração de Marilia | Marilia, Brasil, Marília, São Paulo
  - Centro Avançado de Pesquisa para Diagnóstico - CAPED, Ribeirão Preto, São Paulo
  - Hospital PUC-Campinas | Centro de Pesquisa Clínica Sao Lucas, São Paulo, São Paulo
  - IMC - Instituto de Moléstias Cardiovasculares Tatui, Tatuí, São Paulo
  - Santa Casa de Misericórdia de Votuporanga, Votuporanga, São Paulo
  - Eurolatino Pesquisas Medicas | Uberlandia, MG, Minas Gerais
- Bulgaria (20):
  - Ambulatory facility for specialized outpatient medical care, Burgas
  - MHAT Haskovo, Haskovo
  - MHAT Zdrave, Pazardzhik
  - Multiprofile Hospital for Active Treatment Sveti Georgi OOD, Pernik - Department of Cardiology, Pernik
  - Medical Center Medconsult Pleven, Pleven
  - Medical centre Hipokrat - N EOOD, Plovdiv
  - Multiprofile Hospital for Active Treatment Medline | Cardiology Department, Plovdiv
  - Multiprofile Hospital for Active Treatment Sveta Karidad | Cardiology Department, Plovdiv
  - Multiprofile Hospital for Active Treatment | Shumen - First Department of Internal Medicine, Shumen
  - MHAT Hadzhi Dimitar, Sliven
  - Second Medical Center Sofia EOOD, Sofia
  - Multiprofile Hospital for Active Treatment Knyaginya Klementina Sofia EAD | Cardiology Department, Sofia
  - NMTH Tzar Boris III, Sofia
  - Multiprofile Hospital for Active Treatment 'National Cardiology Hospital' EAD, Sofia, Sofia
  - Multiprofile Hospital for Active Treatment Sveta Sofia | Internal Diseases Department, Sofia
  - Medical Center Hera, Sofia
  - UMHAT Tsaritsa Joanna-ISUL EAD Sofia, Sofia
  - MHAT Trakia, Stara Zagora
  - Multiprofile Hospital for Active Treatment Dr. Stefan Cherkezov | Cardiology Department, Veliko Tarnovo
  - Multiprofile Hospital for Active Treatment Sveti Panteleymon Yambol | Cardiology Department, Yambol
- Canada (21):
  - Fraser Clinical Trials, Inc., New Westminster, British Columbia
  - St. Boniface Hospital, Winnipeg, Manitoba
  - G.A. Research Associates, Ltd., Moncton, New Brunswick
  - Dalhousie University - Queen Elizabeth II (QEII) Health Sciences Centre - Halifax Infirmary (HI), Halifax, Nova Scotia
  - Brampton Clinical Trials, Brampton, Ontario
  - Cambridge Cardiac Care Centre, Cambridge, Ontario
  - Vizel Cardiac Research, Cambridge, Ontario
  - London Health Sciences Centre (LHSC) - University Hospital, London, Ontario
  - KMH Cardiology Clinics Inc., Mississauga, Ontario
  - North York Diagnostic and Cardiac Centre, North York, Ontario
  - Oakville Cardiovascular Research, Oakville, Ontario
  - Office of Dr. James Cha, MD, Oshawa, Ontario
  - Kawartha Cardiology Clinical Trials, Peterborough, Ontario
  - Corcare, Scarborough Village, Ontario
  - Medicus MFC Inc., Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Women's College Hospital, Toronto, Ontario
  - Centre intégré de santé et de services sociaux de Laval, Hôp, Laval, Quebec
  - Clinique Sante Cardio MC, Montreal, Quebec
  - Centre Hospitalier de l'Université de Montréal-CHUM, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
- China (45):
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hosp. Sun Yat-Sen Univ., Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou University of TCM, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - Hainan Provincial People's Hospital, Haikou, Hainan
  - Hainan Third People's Hospital (Province Nongken Sanya Hopt), Sanya, Hainan
  - The First Hospital of Hebei Medical Univesity, Shijiazhuang, Hebei
  - Daqing Oilfield General Hospital, Daqing, Heilongjiang
  - Xinxiang Central Hospital, Xinxiang, Henan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Changsha Central Hospital, Changsha, Hunan
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - Huai'an First People's Hospital, Nanjing Medical University, Huai'an, Jiangsu
  - The First People's Hospital of Lianyungang, Lianyungang, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical university, Nanjing, Jiangsu
  - NJ Drum Tower Hospital, the Affil Hos of NJ Univ Med School, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nanjing Jiangning Hospital, Nanjing, Jiangsu
  - 1st Affiliated hospital of Soochow University, Suzhou, Jiangsu
  - Jilin Province People's Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - Panjin Liaohe Oilfield Gem Flower Hospital, Panjin, Liaoning
  - Yinchuan No.1 People's Hospital, Yinchuan, Ningxia
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Shaanxi Provincial People's Hospital, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi Sheng
  - Jinan Central Hospital, Jinan, Shandong
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - SichuanAcademyofMedicalSciences&SichuanProvincialPeople'sHos, Chengdu, Sichuan
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - 1st Affiliated Hospital of College Medicine, Zhejiang Univ., Hangzhou, Zhejiang
  - Beijing Anzhen Hospital, Capital Medical University, Beijing
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - Beijing Tsinghua Changgung Hospital, Beijing
  - Shanghai Tongji Hospital of Tongji University, Shanghai
  - Shanghai East Hospital Affiated to Tongji University, Shanghai
  - Tianjin People's Hospital, Tianjin
- Colombia (19):
  - Hospital Alma Mater de Antioquia, Medellín, Antioquia
  - Hospital General de Medellin, Medellín, Antioquia
  - Rodrigo Botero S.A.S, Medellín, Antioquia
  - Sociedad Médica Rionegro SOMER S.A., Rionegro, Antioquia
  - Clínica de la Costa SAS, Baranquilla, Atlántico
  - Corazón IPS S.A.S., Barranquilla, Atlántico
  - IPS Centro Cientifico Asistencial S.A.S, Barranquilla, Atlántico
  - Caja de Compensación Familiar CAFAM, Bogotá, Bogota D.C.
  - Hospital Universitario Mayor-MÉDERI, Bogotá, Bogota D.C.
  - Cardiomet Cequin Sas, Armenia, Quindío Department
  - Instituto del Corazón de Bucaramanga, Bucaramanga, Santander Department
  - Mediservis del Tolima IPS S.A.S, Ibagué, Tolima Department
  - Clínica Imbanaco S.A.S, Cali, Valle del Cauca Department
  - Fundacio del Caribe para la Investigacio Bio-Medica (BIOS), Barranquilla
  - Fundación Cardioinfantil, Bogotá
  - Hospital Universitario de San Ignacio, Bogotá
  - Hospital Universitario Clínica San Rafael, Bogotá
  - Hospital San Vicente Fundación, Medellín
  - Clinica Cardio VID, Medellín
- Czechia (23):
  - Fakultní nemocnice Brno - Interní kardiologická klinika, Brno, South Moravian
  - Kardiologie MUDr. Libor Nechvatal s.r.o., Brno
  - Kardiologicka ambulance Brno s.r.o., Brno
  - Kardio Chlumec s.r.o.- Kardiologicka ambulance, Chlumec nad Cidlinou
  - Kardiologicka ambulance, Český Krumlov
  - Poliklinika Dolní Brežany, Dolní Břežany
  - Fakultní Nemocnice Hradec Kralové, Hradec Králové
  - Kromerizska nemocnice a.s., Kroměříž
  - LUNACOR, Centrum pro choroby srdce a cev, Kroměříž
  - Krajska Nemocnice Liberec, Liberec
  - KardioBusak s.r.o., Louny
  - Fakultni nemocnice Plzen, Pilsen
  - Kardiologicka a interni ambulance, Písek
  - Polabska zdravotni, s.r.o., Poděbrady
  - Všeobecná fakultní nemocnice v Praze - II. interní klinika - klinika kardiologie a angiologie, Prague
  - Institut Klinicke a Experimentalni Mediciny, Prague
  - Fakultní nemocnice v Motole, Prague
  - Ustredni vojenska nemocnice Praha, Prague
  - Affidea Praha s.r.o - Kardiologie, Praha 11 - Chodov
  - Kardio s.r.o., Třebíč
  - Nemocnice Podlesi, Třinec
  - Angiocor s.r.o., Zlín
  - Nemocnice Znojmo, Znojmo
- Denmark (9):
  - Aarhus Universitetshospital - Børn og Unge, Århus N
  - Sydvestjysk Sygehus Esbjerg | Kardiologisk Forskningsenhed, Esbjerg
  - Capital Region | Gentofte Hospital - Cardiology Research, Hellerup
  - Capital Region | Herlev Hospital - Heart Disease Department, Herlev
  - Region Midtjylland | Regionshospitalet Godstrup - Clinic for Heart Research, Herning
  - Region Sjælland | Holbaek Sygehus - Cardiology department, Holbæk
  - Hvidovre Hospital - Hjertesygdomme, Hvidovre
  - Regionshospitalet Randers - Medicinsk afdeling, Randers
  - Odense University Hospital | Svendborg Hospital - Cardiovascular Research Unit, Svendborg
- Finland (3):
  - HUS Jorvin sairaala, Espoo
  - Tampereen yliopistollinen sairaala, Tampere
  - Turun yliopistollinen keskussairaala, Turku
- Germany (7):
  - Herzklinik Ulm GbR, Ulm, Baden-Wurttemberg
  - Klinikum der Universität Würzburg, Würzburg, Bavaria
  - Medizinische Hochschule Hannover (MHH), Hanover, Lower Saxony
  - Städt. Kliniken Bielefeld gGmbH, Bielefeld, North Rhine-Westphalia
  - Sana-Klinikum Remscheid GmbH, Remscheid, North Rhine-Westphalia
  - Forschungszentrum Ruhr | KliFoCenter GmbH, Witten, North Rhine-Westphalia
  - Universitätsklinikum Hamburg Eppendorf (UKE), Hamburg
- Greece (12):
  - KAT General Hospital of Athens, Kifissia, Attica
  - University General Hospital of Alexandroupoli, Alexandroupoli
  - General Hosp of Athens "Korgialenio-Benakeio" RCH, Ampelokipi - Athens
  - HIPPOKRATION General Hospital of Athens, Athens
  - G. GENNIMATAS General State Hospital of Athens, Athens
  - ALEXANDRA General Hospital of Athens, Athens
  - University General Hospital of Athens "ATTIKON", Chaïdári
  - University General Hospital of Heraklion - Department of Paediatrics, Heraklion
  - University General Hospital of Larissa, Larissa
  - Konstantopoulio General Hospital of Nea Ionia - AGIA OLGA, Nea Ionia
  - University General Hospital of Patras, Pátrai
  - Hippokration General Hospital of Thessaloniki - 3rd Department of Paediatrics, Nephrology Unit', Thessaloniki
- Hong Kong (4):
  - Prince of Wales Hospital, Hong Kong, N.T
  - Princess Margaret Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - Queen Elizabeth Hospital Hong Kong, Hong Kong
- Hungary (18):
  - Cardiomobile Egeszsegugyi Szolgaltato Kft., Balatonfüred
  - Budai Irgalmasrendi Korhaz, Budapest
  - Budapesti Jahn Ferenc Del-pesti Korhaz es Rendelointezet, Budapest
  - University of Semmelweis/ Semmelweis Egyetem, Budapest
  - Eszak-Pesti Centrumkorhaz-Honvedkorhaz, Budapest
  - Budapesti Uzsoki Utcai Kórház, Budapest
  - Bugat Pal Korhaz, Gyöngyös
  - Pharma4Trial Kft., Gyöngyös
  - Csongrad-Csanad Varmegyei Egeszsegugyi Ellato Kozpont Hodmezovasarhelyi Tagintezmeny, Hódmezővásárhely
  - Borsod-Abauj-Zemplen Varmegyei Korhaz es Egyetemi Oktatokorhaz, Miskolc
  - Nagykanizsai Kanizsai Dorottya Korhaz, Nagykanizsa
  - Medifarma-98 Egeszsegugyi, Kereskedelmi es Szolgaltato Kft., Nyíregyháza
  - Coromed Smo Kft, Pécs
  - Da Vinci Maganklinika, Pécs
  - SZTE ÁOK Szent Györgyi Albert Klinikai Kozpont, Szeged
  - Tolna Varmegyei Balassa Janos Korhaz, Szekszárd
  - Csongrad-Csanad Megyei Dr. Bugyi Istvan Korhaz, Szentes
  - Fejer Varmegyei Szent Gyorgy Egyetemi Oktato Korhaz - II. Belgyogyaszat, Székesfehérvár
- India (5):
  - KEM hospital, Berlin, Maharashtra
  - Deenanath Mangeshkar Hospital, Pune, Maharashtra
  - Max Super Speciality Hospital, Saket, New Delhi, National Capital Territory of Delhi
  - Safdarjung Hospital, New Delhi, National Capital Territory of Delhi
  - The Madras Medical Mission (MMM), Chennai, Tamil Nadu
- Israel (14):
  - Assuta Ashdod Public Hospital (R.A), Ashdod
  - Barzilai Ashkelon University Medical Center | Cardiology Department, Ashkelon
  - Rambam Health Corporation, Haifa
  - Bnai Zion Medical Center | Cardiology Department, Haifa
  - Lady Davis Carmel Medical Center, Haifa
  - Hadassah Hebrew University Hospital Ein Kerem, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Health Corporation of Galilee Medical Center, Nahariya
  - Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Health Corporation of the Ziv Medical Center (R.A.), Safed
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
  - Poria Medical Center | Cardiovascular Department, Tiberias
  - Shamir Medical Center (Assaf Harofeh), Ẕerifin
- Italy (22):
  - Azienda Ospedaliero Universitaria Renato Dulbecco, Catanzaro, Calabria
  - Azienda Ospedaliera Universitaria Federico II Di Napoli - DAI Emergenze Cardiovascolari, Medicina Clinica e Dell'Invecchiamento, Napoli, Campania
  - Azienda Unita Sanitaria Locale Di Bologna_Ospedale Maggiore Pizzardi - Medicina A, Bologna, Emilia-Romagna
  - Azienda Ospedaliero-Universitaria Di Bologna IRCCS_Policlinico Sant'Orsola - Medicina Interna Cardiovascolare, Bologna, Emilia-Romagna
  - University Hospital Of Ferrara, Ferrara, Emilia-Romagna
  - Azienda Unita Sanitaria Locale Di Piacenza, Piacenza, Emilia-Romagna
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII - Cardiologia 1, Bergamo, Lombardy
  - Azienda Socio-Sanitaria Territoriale Del Garda, Brescia, Lombardy
  - Azienda Socio Sanitaria Territoriale Degli Spedali Civili Di Brescia - Cardiologia, Brescia, Lombardy
  - Azienda Socio Sanitaria Territoriale Di Cremona, Cremona, Lombardy
  - Centro Cardiologico Monzino S.p.A., Milan, Lombardy
  - ASST di Monza, Monza Brianza, Lombardy
  - IRCCS Fondazione Policlinico San Matteo, Pavia, Lombardy
  - Istituti Clinici Scientifici Maugeri S.p.A, Pavia, Lombardy
  - Humanitas Mirasole S.p.A. - Cardiologia Clinica e Interventistica, Rozzano, Lombardy
  - ASST Sette Laghi_Ospedale Galmarini - Medicina Generale, Tradate, Lombardy
  - Azienda Socio Sanitaria Territoriale Della Brianza _Ospedale di Vimercate - Medicina Interna, Vimercate, Lombardy
  - A.O.U. Maggiore della Carità, Novara, Piedmont
  - Azienda Unita' Sanitaria Locale Toscana Sud Est, Cortona, Tuscany
  - Azienda Ospedaliera Universitaria Senese, Siena, Tuscany
  - A.O. di Perugia_Hospital Santa Maria della Misericordia - S.C. Cardiologia, Perugia, Umbria
  - Azienda Ospedaliera Universitaria Integrata Verona_Borgo Trento - Cardiologia, Verona, Veneto
- Japan (47):
  - Kasugai Municipal Hospital, Kasugai, Aichi-ken
  - TOYOTA Memorial Hospital, Toyota, Aichi-ken
  - Funabashi Municipal Medical Center, Funabashi, Chiba
  - Steel Memorial Yawata Hospital, Kitakyushu, Fukuoka
  - Onga Nakama Medical Association Onga Hospital, Onga-gun, Fukuoka
  - Ogaki Municipal Hospital, Ōgaki, Gifu
  - Shobara Red Cross Hospital, Shōbara, Hiroshima
  - Hyogo Prefectural HarimaHimeji General Medical Center, Himeji, Hyōgo
  - National Hospital Organization Kobe Medical Center, Kobe, Hyōgo
  - Higashi Takarazuka Satoh Hospital, Takarazuka, Hyōgo
  - JA Toride Medical Center, Toride, Ibaraki
  - Public Central Hospital of Matto Ishikawa | Clinical Trial Management Office, Hakusan, Ishikawa-ken
  - National Hospital Organization Kanazawa Medical Center | Clinical Trial Management Office, Kanazawa, Ishikawa-ken
  - Iwate Prefectural Central Hospital, Morioka, Iwate
  - Kagawa Prefectural Central Hospital, Takamatsu, Kagawa-ken
  - Mitoyo General Hospital | Kagawa, Japan, Toyohama-Cho,Kanonji-City, Kagawa-ken
  - Kitasato University Hospital, Sagamihara, Kanagawa
  - Sagamihara Kyodo Hospital, Sagamihara, Kanagawa
  - Japan Red Cross Society Azumino Hospital, Azumino, Nagano
  - National Hospital Organization Shinshu Ueda Medical Center, Ueda, Nagano
  - R.I.A.C Naha City Hospital, Naha, Okinawa
  - Kishiwada Tokushukai Hospital, Kishiwada, Osaka
  - Takatsuki Red Cross Hospital, Takatsuki, Osaka
  - Ageo Central General Hospital, Ageo, Saitama
  - Kawaguchi Cardiovascular and Respiratory Hospital, Kawaguchi, Saitama
  - Saitama Sekishinkai Hospital, Sayama, Saitama
  - National Hospital Organization Hamada Medical Center, Hamada, Shimane
  - Nishiarai Heart Central Clinic, Adachi-ku, Tokyo
  - Minamino Cardiovascular Hospital, Hachiōji, Tokyo
  - National Hospital Organization Tokyo Medical Center, Meguro-ku, Tokyo
  - Toho University Omori Medical Center, Ōta-ku, Tokyo
  - Japan Organization of Occupational Health and Safety Sanin Rosai Hospital, Yonago, Tottori
  - National Hospital Organization Iwakuni Clinical Center, Iwakuni, Yamaguchi
  - JCHO Shimonoseki Medical Center, Shimonoseki, Yamaguchi
  - Fukuoka University Nishijin Hospital, Fukuoka
  - Gifu Prefectural General Medical Center, Gifu
  - National Hospital Organization Kumamoto Medical Center, Kumamoto
  - Kumamoto University Hospital, Kumamoto
  - Miyazaki Medical Association Hospital, Miyazaki
  - Shinrakuen Hospital, Niigata
  - The Sakakibara Heart Institute of Okayama, Okayama
  - Osaka Police Hospital | Clinical Research and Trial Center, Osaka
  - Osaka General Medical Center, Osaka
  - Social Corporation Keigakukai Minamiosaka Hospital, Osaka
  - Oita Prefectural Hospital, Ōita
  - Toyama University Hospital, Toyama
  - Seiyu Memorial Hospital, Wakayama
- Latvia (7):
  - Daugavpils Regional Hospital, Daugavpils
  - Jelgava Outpatient Clinic, Jelgava
  - Liepaja Regional Hospital, Liepāja
  - 1st Riga Clinical Hospital, Riga
  - P. Stradins Clinical University Hospital, Riga
  - GK Neiroklinika, Riga
  - Gita Rancane - cardiology private practice, Ventspils
- Lithuania (7):
  - UAB "Klinikiniai sprendimai" Alytus, Alytus
  - LUHS Kauno Hospital (Laisves ave.), Kaunas
  - LUHS Kauno Hospital (Josvainiu str.), Kaunas
  - Saules family medicine center, Kaunas
  - Klaipedos Jurininku Ligonine, Klaipėda
  - Siauliai Republican hospital, Šiauliai
  - Vilnius University Hospital Santaros Klinikos, Vilnius
- Malaysia (7):
  - Gleneagles Penang Medical Center, George Town
  - Institute Jantung Negara, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Sultan Idris Shah Serdang (Hospital Serdang), Kuala Selangor
  - Hospital Raja Permaisuri Bainun, Perak
  - Hospital Pulau Pinang, Pulau Pinang
  - Sarawak Heart Centre, Sarawak
- Mexico (9):
  - Centro de Investigación Médica Dr. Alberto Bazzoni SA de CV, Torreón, Coahuila
  - Hospital General de Acapulco, Acapulco de Juárez, Guerrero
  - Consultorio de Medicina Especializada del Sector Privado, Guadalajara, Jalisco
  - Fundación de Atencion e Investigacion Medica Lindavista SC, Alcaldia Gustavo A. Madero, Mexico City
  - Hospital de Jesús, Alcaldía Cuauhtemoc, Mexico City
  - Centro de Estudios Clinicos de Queretaro S. C. (CECLIQ), Querétaro City, Querétaro
  - Hospital Ángeles de Xalapa, Xalapa, Veracruz
  - Hospital Cardiologica Aguascalientes, Aguascalientes
  - Centro de Investigacion y Atencion Integral Durango S.C., Durango
- Netherlands (13):
  - Catharina Ziekenhuis, Eindhoven, North Brabant
  - Ziekenhuis Groep Twente, Almelo
  - Deventer Ziekenhuis, Deventer
  - Slingeland Ziekenhuis, Doetinchem
  - Ziekenhuis Gelderse Vallei, Ede
  - Universitair Medisch Centrum Groningen, Groningen
  - Ziekenhuis St. Jansdal, Harderwijk
  - Tergooiziekenhuizen-Blaricum, Hilversum
  - Maastricht UMC, Maastricht
  - Isala Meppel, Meppel
  - Antonius Ziekenhuis Sneek, Sneek
  - ETZ TweeSteden Ziekenhuis (vh Maria Ziekenhuis), Tilburg
  - Maxima Medisch Centrum, locatie Veldhoven, Veldhoven
- New Zealand (7):
  - University of Auckland, Auckland
  - Christchurch Heart Institute, Christchurch
  - Dunedin Hospital, Dunedin
  - P3 Research Ltd Tauranga, Hawkes Bay
  - Hutt Hospital, Lower Hutt
  - Nelson Hospital, Nelson
  - P3 Research, Tauranga
- Poland (15):
  - KLIMED Marek Klimkiewicz, Bialystok
  - MICS Centrum Medyczne Bydgoszcz, Bydgoszcz
  - Uniwersyteckie Centrum Medycyny Morskiej i Tropikalnej, Gdynia
  - Samodzielny Publiczny Specjalistyczny Szpital Zachodni im. sw. Jana Pawla II, Grodzisk Mazowiecki
  - CLINICAL MEDICAL RESEARCH Sp. z o. o., Katowice
  - Unicardia Specjalistyczne Centrum Leczenia Ch.Serca i Naczyn, Krakow
  - IMEDICA Centrum Medyczne, Lublin
  - NZOZ "Twoja Przychodnia" Sp. z o.o., Lublin
  - Zechowicz Medeusz-Plus Lekarska Spolka Partnerska, Olsztyn
  - Oswiecimskie Centrum Badan Klinicznych Medicome Sp. z o.o., Oświęcim
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Poznan
  - Szpital Specjalistyczny SPZOZ, Puławy
  - NZOZ Pro-Cordis Sopockie Centrum Badan Kardiologicznych, Sopot
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin
  - Gessek Jacek Prywatny Gabinet Lekarski, Torun
- Portugal (12):
  - Hospital da Senhora da Oliveira | Clinical Research Department, Guimaraes, Braga, Braga District
  - Centro Hospitalar Universitario Cova de Beira | Clinical Research Department, Covilha, Castelo Branco District
  - Hospital Pedro Hispano | Clinical Research Center, Matosinhos Municipality, Porto District
  - Luz Saude | Hospital da Luz Setubal - Clinical Research Department, Setúbal, Setúbal District
  - Hospital Prof. Dr. Fernando Fonseca, Amadora
  - BlueClinical | Centro Hospitalar Baixo Vouga - Unidade Aveiro - Gabinete de Ensaios Clinicos, Aveiro
  - Unidade Local de Saúde de Coimbra, E.P.E. - Cardiology Department - Research Unit, Coimbra
  - ULSG - Unidade Local de Saude da Guarda, Guarda
  - Centro Hospitalar de Leiria | Santo Andre Hospital - Research Center, Leiria
  - Unidade Local De Saúde De Lisboa Ocidental E.P.E., Lisbon
  - Luz Saude | Hospital da Luz Lisboa - Centro de Investigacao Clinica, Lisbon
  - Centro Hospitalar Universitario do Porto, Porto
- Romania (15):
  - CMI. Dr. Podoleanu Cristian, Târgu Mureş, Mureș County
  - Spitalul Clinic Municipal de Urgenta "Timisoara", Timișoara, Timiș County
  - Municipal Clinical Emergency Hospital of Timisoara, Timișoara, Timiș County
  - Sp. Judetean de Urgenta Dr. Constantin Opris Baia Mare, Baia Mare
  - S.C Thera Card S.R.L, Brasov
  - Emergency County Hospital, Braila, Brăila
  - Emergency Institute for Cardiovascular Diseases, Bucharest
  - Spitalul Universitar de Urgenta Bucuresti, Bucharest
  - Spitalul Clinic de Urgenta "Sf. Pantelimon", Bucharest
  - Spitalul Clinic Judetean De Urgenta Craiova, Craiova Dolj
  - Sf. Ap. Andrei Emergency Clinical County Hospital Galati, Galati
  - S.C. CARDIOMED S.R.L. Iasi, Iași
  - S.C. Sal Med SRL, Piteşti
  - S.C. Cardio Med S.R.L., Târgu Mureş
  - Institutul De Boli Cardiovasculare Timisoara, Timișoara
- Russia (28):
  - SBHI of Sverdlovsk Region Aramil City Hospital, Aramil
  - First City Clinical Hospital n.a. E.E. Volosevich, Arkhangelsk
  - Altai Regional Cardiological Dispensary, Barnaul
  - SBEI "Chita State Medical Academy", Chita
  - Izhevsk City Clinical Hospital #9, Izhevsk
  - Kazan Federal University, Kazan'
  - Clinical Diagnostic Center, Kazan'
  - Sci-Res. Institute of Complex Cardiovascular Disorders, Kemerovo
  - Center of cardiology and neurology, Kirov
  - Research center of therapy and prophylactic medicine, Moscow
  - City Clinical Hospital #29 n.a. N.E. Bauman - Clinical-Diagnostic dept, Moscow
  - City clinical hospital n.a. V.V. Vinogradov, Moscow
  - Moscow State University n.a. M.V. Lomonosov, Moscow
  - Russian Clinical and Research Center of Gerontology, Moscow
  - State Novosibirsk Regional Clinical Hospital, Novosibirsk
  - Omsk Region "Clinical Health Unit No. 9", Omsk
  - Penza Regional Clinical Hospital n.a. N.N. Burdenko, Penza
  - Perm Regional Hospital for War Veterans, Perm
  - Rostov-on-Don Emergency Clinical Hospital, Rostov-on-Don
  - SBI of the Ryazan region "Regional clinical hospital", Ryazan
  - Scien. Res. Inst. of Emergency Care n.a. I.I. Dzhanelidze, Saint Petersburg
  - St. Petersburg Clinical Hospital of RAS, Saint Petersburg
  - LLC Astarta, Saint Petersburg
  - Samara Regional Clinical Cardiology Dispensary n.a. Polyakov, Samara
  - Clinical Hospital #3 n.a. S.R. Mirotvortsev, Saratov
  - Scientific Research Institute of Cardiology, Tomsk
  - Tomsk Regional Clinical Hospital, Tomsk
  - Sverdlovsk Regional Clinical Hospital #1, Yekaterinburg
- Slovakia (19):
  - Stredoslovensky ustav srdcovych a cievnych chorob, a.s., Banská Bystrica
  - ALIAN s.r.o., Bardejov
  - Nemocnica svateho Michala, a.s., Bratislava
  - Univerzitna nemocnica Bratislava, Nemocnica Stare Mesto, Bratislava
  - Narodny ustav srdcovych a cievnych chorob, a.s, Bratislava
  - Centrum interv. neuroradiologie a endovaskularnej liecby, Bratislava
  - Kardiosanus | Bratislava, Slovakia, Bratislava
  - Nemocnica s poliklinikou Brezno, n.o., Brezno
  - Dolnooravska nemocnica s poliklinikou L. Nadasi Jegeho, Dolný Kubín
  - JG-COR s.r.o., Košice
  - Medical Group Kosice s.r.o. | Kosice, Slovakia, Košice
  - KARDIO-ANGIO s.r.o., Levice
  - KardioMed s.r.o., Lučenec
  - MEDI M&M, s.r.o., Moldava nad Bodvou
  - Kardiocentrum Nitra | Cardiology Clinic - Outpatient Department, Nitra
  - KARDIOMED NZ s.r.o., Nové Zámky
  - MEDISPOL s.r.o., Prešov
  - COR, s.r.o, Šahy
  - Medivasa s.r.o., Žilina
- South Korea (10):
  - Yonsei University Wonju Christian Hospital, Wŏnju, Gang''weondo
  - Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggido
  - Bundang Cha Hospital, Seongnam-si, Gyeonggido
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Dong-A University Hospital, Busan
  - Pusan National University Hospital, Busan
  - Chung Nam National University Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
- Spain (23):
  - Complejo Hospitalario Universitario de Ferrol | Hospital Naval - Unidad de Hipertensión Arterial, Ferrol, A Coruña
  - Hospital Vega Baja De Orihuela - Medicina Interna, San Bartolomé, Alicante
  - Hospital Santa María del Puerto - Medicina Interna, El Puerto de Santa María, Cádiz
  - Hospital Virgen del Camino - Medicina Interna, Sanlúcar de Barrameda, Cádiz
  - Hospital Virgen De Las Montanas - Medicina Interna, Villamartín, Cádiz
  - Hospital Universitario de Gran Canaria Dr. Negrin - Cardiologia, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Virgen De La Victoria - Cardiologia, Málaga, Málaga
  - Hospital Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Alta Resolucion de Utrera - Cardiologia, Utrera, Sevilla
  - Instituto Medico Quirurgico San Rafael S.A. - Cardiologia, A Coruña
  - Hospital del Mar, Barcelona
  - Ciutat Sanitaria i Universitaria de la Vall d'Hebron, Barcelona
  - Hospital Universitari de Bellvitge (HUB), Barcelona
  - Hospital Universitario Virgen De Las Nieves - Cardiologia, Granada
  - Hospital Universitari Arnau De Vilanova De La Gerencia Territorial De Lleida - Medicina Interna, Lleida
  - Hospital Universitario La Zarzuela - Cardiologia, Madrid
  - Hospital Ramón y Cajal | Medicina Interna, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen de Valme - Medicina Interna, Seville
  - Hospital Clinico Universitario de Valencia (CHUV), Valencia
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario Y Politecnico La Fe - Cardiologia, Valencia
  - Hospital de Manises - Medicina Interna, Valencia
- Taiwan (8):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Kaohsiung
  - Changhua Christian Hospital, Changhua
  - Mackay Memorial Hospital - Hsinchu Branch, Hsinchu
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital at Linkou, Taoyuan District
- Turkey (Türkiye) (13):
  - Afyonkarahisar Saglik Bilimleri Universitesi, Afyonkarahisar
  - Saglik Bilimleri Universitesi Antalya EA Hastanesi, Antalya
  - Trakya Univ. Tip Fak., Edirne
  - Eskisehir Osmangazi Universitesi Tip Fakultesi, Eskişehir
  - Istanbul Universitesi Cerrahpasa-Cerrahpasa Tip Fakultesi, Istanbul
  - Istanbul Universitesi Kardiyoloji Enstitusu, Istanbul
  - Istanbul Mehmet Akif Ersoy Gogus Kalp Damar Cerrahisi E.A.H., Istanbul
  - Dokuz Eylul Universitesi Tip Fakultesi, Izmir
  - Erciyes Universitesi Tip Fakultesi, Kayseri
  - Kocaeli Universitesi Tip Fakultesi, Kocaeli
  - Necmettin Erbakan Universitesi Meram Tip Fakultesi Hastanesi, Konya
  - Kutahya Saglik Bilimleri Uni. Evliya Celebi Egitim ve Arasti, Kütahya
  - Mersin Universitesi Tip Fakultesi, Mersin
- Ukraine (21):
  - MNPE "Cherkasy Regional Cardiology Center" - Department of Coronary Heart Disease and Non-Coronary Myocardial Diseases, Cherkasy
  - Clinical Emergency Hospital" of Dnipro City Council - Department of Cardiology, Dnipro
  - National Institute of Therapy L.T.Maloyi, Department of Chronic Non-Communicable Diseases, Kharkiv
  - Regional Dispensary of Radiation Protection of Population - Cardiology Department, Kharkiv
  - MNPE "City Clinical Hospital No. 8" of the Kharkiv City Council, Cardiology Department No. 2, Kharkiv
  - Municipal Non-Profit Enterprise "Kyiv City Clinical Hospital No. 1" - Department of Cardiology, Kiev
  - Medical Center "Medbud" - Treatment and prophylactic department, Kyiv
  - National Scientific Center Institute of Cardiology named M.D. Strazhesko of the NAMSU - Department of Cardiac Arrhythmias, Kyiv
  - National Scientific Center Institute of Cardiology named M.D. Strazhesko of the NAMSU - Department of Heart Failure, Kyiv
  - National Scientific Center Institute of Cardiology named M.D. Strazhesko of the NAMSU - Department of Hypertension, Kyiv
  - LLC "Medical Center "Consilium Medical", Clinical and Consultative Departmen 1, Kyiv
  - Railway Clinical Hospital #2, Kyiv
  - Lviv Regional Clinical Treatment and Diagnostic Cardiology Center, consulting polyclinic, Lviv
  - Poltava Regional Clinical Hospital. M.V. Sklifosovsky, Cardiology Department, Poltava
  - Zakarpatsky Oblasnyi Kardiologichnyi Dyspanser, Infarction department, Uzhhorod
  - Vinnytsia Regional Clinical Hospital, Clinical Cardiology Department, Vinnytsia
  - Vinnytsia City Clinical Hospital #1, Therapeutic Department, Vinnytsia
  - Regional Medical Center for Cardiovascular Diseases-Heart failure department, Zaporizhzhia
  - Zaporizhia Municipal Clinical Hospital No.10, Cardiology Department, Zaporizhzhya
  - Zaporizhzhya City Emergency Care Hospital, Cardiology Department, Zaporizhzhya
  - Hospital No. 1 of the Zhytomyr City - consulting and treatment department Scientific and research center, Zhytomyr
- United Kingdom (14):
  - Royal Bournemouth General Hospital, Bournemouth, Dorset
  - Poole Hospital NHS Trust, Poole, Dorset
  - Queen Elizabeth University Hospital, Glasgow, Glasgow City
  - North Hampshire Hospital, Basingstoke, Hampshire
  - Lister Hospital, Stevenage, Hertfordshire
  - Blackpool Victoria Hospital, Blackpool, Lancashire
  - University Hospitals Leicester, Leicester, Leicestershire
  - Wansbeck General Hospital, Ashington, Northumberland
  - Dudley Group NHS Foundation Trust ¦Russells Hall Hopsital - Oncology, Dudley, West Midlands
  - University Hospitals Sussex NHS Foundation Trust | St Richard's Hospital - Cardiology services, Chichester, West Sussex
  - Hull University Teaching Hospitals NHS Trust | Castle Hill Hospital - Cardiology, Cottingham
  - NHS Greater Glasgow and Clyde | Glasgow Royal Infirmary |Glasgow Research Facility - Cardiology, Glasgow
  - Manchester Royal Infirmary, Manchester
  - Great Western Hospital, Swindon

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Result] Bhatt AS, Chatur S, Claggett BL, Lay-Flurrie J, Viswanathan P, Vardeny O, Kosiborod MN, Sharma K, Solomon SD, Vaduganathan M. Gamified Behavioral Science Intervention to Enhance Trial Enrollment: An Embedded Study Within the FINEARTS-HF Trial. JACC Heart Fail. 2024 Nov;12(11):1939-1941. doi: 10.1016/j.jchf.2024.05.002. Epub 2024 May 11. No abstract available. PMID 38944793
- [Result] Jhund PS, Talebi A, Henderson AD, Claggett BL, Vaduganathan M, Desai AS, Lam CSP, Pitt B, Senni M, Shah SJ, Voors AA, Zannad F, Solomon SD, McMurray JJV. Mineralocorticoid receptor antagonists in heart failure: an individual patient level meta-analysis. Lancet. 2024 Sep 21;404(10458):1119-1131. doi: 10.1016/S0140-6736(24)01733-1. Epub 2024 Sep 1. PMID 39232490
- [Result] Kondo T, Henderson AD, Docherty KF, Jhund PS, Vaduganathan M, Solomon SD, McMurray JJV. Why Have We Not Been Able to Demonstrate Reduced Mortality in Patients With HFmrEF/HFpEF? J Am Coll Cardiol. 2024 Nov 26;84(22):2233-2240. doi: 10.1016/j.jacc.2024.08.033. Epub 2024 Sep 1. PMID 39217560
- [Result] Ostrominski JW, Aggarwal R, Claggett BL, Kulac IJ, Desai AS, Jhund PS, Lam CSP, Pitt B, Senni M, Shah SJ, Voors AA, Zannad F, Lay-Flurrie J, Viswanathan P, McMurray JJV, Solomon SD, Vaduganathan M. Generalizability of the Spectrum of Kidney Risk in the FINEARTS-HF Trial to U.S. Adults With Heart Failure. J Card Fail. 2024 Sep;30(9):1170-1174. doi: 10.1016/j.cardfail.2024.04.015. Epub 2024 May 11. No abstract available. PMID 38740173
- [Result] Ostrominski JW, Claggett BL, Miao ZM, Mc Causland FR, Anand IS, Desai AS, Jhund PS, Lam CSP, Pfeffer MA, Pitt B, Zannad F, Zile MR, Bomfim Wirtz A, Lay-Flurrie J, Viswanathan P, McMurray JJV, Solomon SD, Vaduganathan M. Cardiovascular-Kidney-Metabolic Overlap in Heart Failure With Mildly Reduced or Preserved Ejection Fraction: A Trial-Level Analysis. J Am Coll Cardiol. 2024 Jul 9;84(2):223-228. doi: 10.1016/j.jacc.2024.05.005. Epub 2024 May 12. No abstract available. PMID 38744407
- [Result] Solomon SD, McMurray JJV, Vaduganathan M, Claggett B, Jhund PS, Desai AS, Henderson AD, Lam CSP, Pitt B, Senni M, Shah SJ, Voors AA, Zannad F, Abidin IZ, Alcocer-Gamba MA, Atherton JJ, Bauersachs J, Chang-Sheng M, Chiang CE, Chioncel O, Chopra V, Comin-Colet J, Filippatos G, Fonseca C, Gajos G, Goland S, Goncalvesova E, Kang S, Katova T, Kosiborod MN, Latkovskis G, Lee AP, Linssen GCM, Llamas-Esperon G, Mareev V, Martinez FA, Melenovsky V, Merkely B, Nodari S, Petrie MC, Saldarriaga CI, Saraiva JFK, Sato N, Schou M, Sharma K, Troughton R, Udell JA, Ukkonen H, Vardeny O, Verma S, von Lewinski D, Voronkov L, Yilmaz MB, Zieroth S, Lay-Flurrie J, van Gameren I, Amarante F, Kolkhof P, Viswanathan P; FINEARTS-HF Committees and Investigators. Finerenone in Heart Failure with Mildly Reduced or Preserved Ejection Fraction. N Engl J Med. 2024 Oct 24;391(16):1475-1485. doi: 10.1056/NEJMoa2407107. Epub 2024 Sep 1. PMID 39225278
- [Result] Solomon SD, Ostrominski JW, Vaduganathan M, Claggett B, Jhund PS, Desai AS, Lam CSP, Pitt B, Senni M, Shah SJ, Voors AA, Zannad F, Abidin IZ, Alcocer-Gamba MA, Atherton JJ, Bauersachs J, Ma CS, Chiang CE, Chioncel O, Chopra V, Comin-Colet J, Filippatos G, Fonseca C, Gajos G, Goland S, Goncalvesova E, Kang SM, Katova T, Kosiborod MN, Latkovskis G, Lee AP, Linssen GCM, Llamas-Esperon G, Mareev V, Martinez FA, Melenovsky V, Merkely B, Nodari S, Petrie MC, Saldarriaga CI, Saraiva JFK, Sato N, Schou M, Sharma K, Troughton R, Udell JA, Ukkonen H, Vardeny O, Verma S, von Lewinski D, Voronkov LG, Yilmaz MB, Zieroth S, Lay-Flurrie J, van Gameren I, Amarante F, Viswanathan P, McMurray JJV. Baseline characteristics of patients with heart failure with mildly reduced or preserved ejection fraction: The FINEARTS-HF trial. Eur J Heart Fail. 2024 Jun;26(6):1334-1346. doi: 10.1002/ejhf.3266. Epub 2024 May 11. PMID 38733212
- [Result] Vaduganathan M, Claggett BL, Lam CSP, Pitt B, Senni M, Shah SJ, Voors AA, Zannad F, Desai AS, Jhund PS, Viswanathan P, Bomfim Wirtz A, Schloemer P, Lay-Flurrie J, McMurray JJV, Solomon SD. Finerenone in patients with heart failure with mildly reduced or preserved ejection fraction: Rationale and design of the FINEARTS-HF trial. Eur J Heart Fail. 2024 Jun;26(6):1324-1333. doi: 10.1002/ejhf.3253. Epub 2024 May 14. PMID 38742248
- [Result] Vaduganathan M, Filippatos G, Claggett BL, Desai AS, Jhund PS, Henderson A, Brinker M, Kolkhof P, Schloemer P, Lay-Flurrie J, Viswanathan P, Lam CSP, Senni M, Shah SJ, Voors AA, Zannad F, Rossing P, Ruilope LM, Anker SD, Pitt B, Agarwal R, McMurray JJV, Solomon SD. Finerenone in heart failure and chronic kidney disease with type 2 diabetes: FINE-HEART pooled analysis of cardiovascular, kidney and mortality outcomes. Nat Med. 2024 Dec;30(12):3758-3764. doi: 10.1038/s41591-024-03264-4. Epub 2024 Sep 1. PMID 39218030
- [Result] Vaduganathan M, Neuen BL, McCausland F, Jhund PS, Docherty KF, McMurray JJV, Solomon SD. Why Has it Been Challenging to Modify Kidney Disease Progression in Patients With Heart Failure? J Am Coll Cardiol. 2024 Nov 26;84(22):2241-2245. doi: 10.1016/j.jacc.2024.08.034. Epub 2024 Sep 1. No abstract available. PMID 39217561
- [Derived] Chimura M, Henderson AD, Jhund PS, Claggett BL, Desai AS, Filippatos G, Gajos G, Brinker M, Amarante F, Lay-Flurrie J, Rohwedder K, Lam CSP, Sato N, Senni M, Voors AA, Zannad F, Yilmaz MB, Pitt B, Vaduganathan M, Solomon SD, McMurray JJV. Efficacy and Safety of the Kidney Function-Based Finerenone Dosing Strategy Used in FINEARTS-HF. JACC Heart Fail. 2026 Feb 2:102938. doi: 10.1016/j.jchf.2026.102938. Online ahead of print. PMID 41642173
- [Derived] Butt JH, Henderson AD, Jhund PS, Claggett BL, Desai AS, Borentain M, Rohwedder K, Dayoub R, De Sanctis Y, Lam CSP, Senni M, Shah SJ, Voors AA, Bauersachs J, Fonseca C, Linssen GCM, Petrie MC, Schou M, Verma S, Zannad F, Pitt B, Vaduganathan M, Solomon SD, McMurray JJV. Finerenone, Liver Biomarkers, and Heart Failure With Mildly Reduced/Preserved Ejection Fraction: An Analysis of FINEARTS-HF. Circ Heart Fail. 2026 Jan 29:e013201. doi: 10.1161/CIRCHEARTFAILURE.125.013201. Online ahead of print. PMID 41608790
- [Derived] Foa A, Vaduganathan M, Claggett BL, Desai AS, Jhund PS, Henderson AD, Chatur S, Amarante F, Hofmeister L, Horvat-Broecker A, Kuhls S, Lam CSP, Senni M, Shah SJ, Voors AA, Zannad F, Pitt B, McMurray JJV, Solomon SD. Finerenone-Related Risk of Hypotension in Heart Failure With Mildly Reduced or Preserved Ejection Fraction. JACC Heart Fail. 2025 Dec 6:102779. doi: 10.1016/j.jchf.2025.102779. Online ahead of print. PMID 41364043
- [Derived] Ostrominski JW, Claggett BL, Desai AS, Jhund PS, Lam CSP, Senni M, Shah SJ, Voors AA, Zannad F, Pitt B, Rohwedder K, Brinker M, Schloemer P, McMurray JJV, Solomon SD, Vaduganathan M. Finerenone according to insulin resistance in heart failure: Insights from the FINEARTS-HF trial. Eur J Heart Fail. 2025 Dec;27(12):2788-2799. doi: 10.1002/ejhf.70034. Epub 2025 Sep 8. PMID 40916719
- [Derived] Lu H, Claggett BL, Vaduganathan M, Desai AS, Jhund PS, Voors AA, Senni M, Zannad F, Pitt B, Shah SJ, Lam CSP, Scheerer MF, Scalise A, Mueller K, Berger M, Goea L, McMurray JJV, Solomon SD. Temporal Changes in Biomarkers, Functional Status, and Quality of Life Prior to Adverse Clinical Outcomes in Heart Failure With Mildly Reduced or Preserved Ejection Fraction. JACC Heart Fail. 2025 Oct;13(10):102590. doi: 10.1016/j.jchf.2025.102590. Epub 2025 Aug 25. PMID 40857999
- [Derived] Chimura M, Jhund PS, Henderson AD, Yang M, Claggett BL, Desai AS, Rohwedder K, Lage A, Scalise A, Mueller K, Schou M, Lam CSP, Senni M, Voors AA, Zannad F, Pitt B, Vaduganathan M, Solomon SD, McMurray JJV. Efficacy and Tolerability of Finerenone According to the Use and Dosage of Diuretics: A Prespecified Analysis of the FINEARTS-HF Randomized Clinical Trial. JAMA Cardiol. 2025 Aug 13;10(10):979-89. doi: 10.1001/jamacardio.2025.2551. Online ahead of print. PMID 40802267
- [Derived] Butt JH, Jhund PS, Henderson AD, Claggett BL, Chiang CE, Linssen GCM, Saldarriaga CI, Saraiva JFK, Sato N, Schou M, von Lewinski D, Lay-Flurrie J, Scalise A, Rohwedder K, Desai AS, Lam CSP, Senni M, Shah SJ, Zannad F, Pitt B, Vaduganathan M, Solomon SD, McMurray JJV. Finerenone According to Frailty in Heart Failure: A Prespecified Analysis of the FINEARTS-HF Randomized Clinical Trial. JAMA Cardiol. 2025 Aug 1;10(8):829-840. doi: 10.1001/jamacardio.2025.1775. PMID 40531488
- [Derived] Pabon MA, Vardeny O, Vaduganathan M, Desai AS, Claggett BL, Kulac IJ, Jhund PS, Lam CSP, Senni M, Shah SJ, Voors AA, Zannad F, Pitt B, Saldarriaga CI, Petrie MC, Merkely B, Borentain M, Mueller K, Viswanathan P, Amarante F, Morris A, McMurray JJV, Solomon SD. Finerenone in Heart Failure With Improved Ejection Fraction: The FINEARTS-HF Randomized Clinical Trial. JAMA Cardiol. 2025 Jul 1;10(7):740-745. doi: 10.1001/jamacardio.2025.1101. PMID 40397470
- [Derived] Chimura M, Yang M, Henderson AD, Jhund PS, Docherty KF, Claggett BL, Desai AS, Filippatos G, Gajos G, Mueller K, Glasauer A, Rohwedder K, Viswanathan P, Lam CSP, Sato N, Senni M, Voors AA, Zannad F, Yilmaz MB, Pitt B, Vaduganathan M, Solomon SD, McMurray JJV; FINEARTS-HF Committees and Investigators. Anaemia in patients with heart failure and mildly reduced or preserved ejection fraction: A prespecified analysis of the FINEARTS-HF trial. Eur J Heart Fail. 2025 Nov;27(11):2301-2312. doi: 10.1002/ejhf.3682. Epub 2025 May 16. PMID 40377177
- [Derived] Kondo T, Jhund PS, Henderson AD, Claggett BL, Desai AS, Brinker M, Lay-Flurrie J, Schloemer P, Viswanathan P, Amarante F, Chiang CE, Filippatos G, Lam CSP, Petrie MC, Senni M, Schou M, Verma S, Voors AA, von Lewinski D, Zannad F, Pitt B, Vaduganathan M, Solomon SD, McMurray JJV. The efficacy of finerenone on hierarchical composite endpoint analysed using win statistics in patients with heart failure and mildly reduced or preserved ejection fraction: A prespecified analysis of FINEARTS-HF. Eur J Heart Fail. 2025 Aug;27(8):1459-1471. doi: 10.1002/ejhf.3669. Epub 2025 Apr 29. PMID 40300840
- [Derived] Ostrominski JW, Vaduganathan M, Claggett BL, Desai AS, Jhund PS, Lam CSP, Senni M, Shah SJ, Voors AA, Zannad F, Pitt B, Borentian M, Rohwedder K, Lay-Flurrie J, Lavagnino MA, McMurray JJV, Solomon SD. Finerenone and NYHA Functional Class in Heart Failure: The FINEARTS-HF Trial. JACC Heart Fail. 2026 Jan;14(1):102440. doi: 10.1016/j.jchf.2025.03.007. Epub 2025 Apr 2. PMID 40232214
- [Derived] Butt JH, Jhund PS, Henderson AD, Claggett BL, Desai AS, Lam CSP, Mueller K, Scheerer MF, Viswanathan P, Senni M, Shah SJ, Voors AA, Zannad F, Pitt B, Vaduganathan M, Solomon SD, McMurray JJV. Finerenone, chronic obstructive pulmonary disease, and heart failure with mildly reduced or preserved ejection fraction: A prespecified analysis of the FINEARTS-HF trial. Eur J Heart Fail. 2025 Aug;27(8):1444-1458. doi: 10.1002/ejhf.3661. Epub 2025 Apr 13. PMID 40222820
- [Derived] Ostrominski JW, Mc Causland FR, Claggett BL, Desai AS, Jhund PS, Lam CSP, Senni M, Shah SJ, Voors AA, Zannad F, Pitt B, Schloemer P, Brinker M, Scheerer MF, McMurray JJV, Solomon SD, Vaduganathan M. Finerenone Across the Spectrum of Kidney Risk in Heart Failure: The FINEARTS-HF Trial. JACC Heart Fail. 2025 Apr 2:102439. doi: 10.1016/j.jchf.2025.03.006. Online ahead of print. PMID 40208137
- [Derived] Desai AS, Jhund PS, Vaduganathan M, Claggett BL, Cunningham JW, Pabon MA, Lam CSP, Senni M, Shah S, Voors AA, Zannad F, Pitt B, Amarante F, Lay-Flurrie J, Scheerer MF, Lage A, McMurray JJV, Solomon SD. Mode of Death in Patients With Heart Failure With Mildly Reduced or Preserved Ejection Fraction: The FINEARTS-HF Randomized Clinical Trial. JAMA Cardiol. 2025 Jul 1;10(7):678-685. doi: 10.1001/jamacardio.2025.0860. PMID 40159247
- [Derived] Matsumoto S, Henderson AD, Jhund PS, Bauersachs J, Chioncel O, Claggett BL, Comin-Colet J, Desai AS, Filippatos G, Lam CSP, Pitt B, Scheerer MF, Lay-Flurrie J, Amarante F, Brinker M, Schou M, Senni M, Shah SJ, Voors AA, Zannad F, Zieroth S, Vaduganathan M, Solomon SD, McMurray JJV. Finerenone and Atrial Fibrillation in Heart Failure: A Secondary Analysis of the FINEARTS-HF Randomized Clinical Trial. JAMA Cardiol. 2025 Jul 1;10(7):696-707. doi: 10.1001/jamacardio.2025.0848. PMID 40156827
- [Derived] McDowell K, Docherty KF, Campbell RT, Henderson AD, Jhund PS, Claggett BL, Desai AS, Lay-Flurrie J, Hofmeister L, Scalise A, Lam CSP, Petrie MC, Schou M, Senni M, Shah SJ, Udell JA, Zannad F, Pitt B, Vaduganathan M, Solomon SD, McMurray JJV. Finerenone for Heart Failure and Risk Estimated by the PREDICT-HFpEF Model: A Secondary Analysis of FINEARTS-HF. JAMA Cardiol. 2025 Jun 1;10(6):535-544. doi: 10.1001/jamacardio.2025.0025. PMID 40042880
- [Derived] Cunningham JW, Chatur S, Claggett BL, Vaduganathan M, Desai AS, Jhund PS, Llamas Esperon G, Lam CSP, Sato N, Senni M, Shah S, Voors A, Zannad F, Pitt B, Zieroth S, Brinker M, Rohwedder K, Kim SY, Lay-Flurrie J, Viswanathan P, McMurray JJV, Solomon SD. Finerenone and Outpatient Worsening Heart Failure With Mildly Reduced or Preserved Ejection Fraction: A Secondary Analysis of the FINEARTS-HF Randomized Clinical Trial. JAMA Cardiol. 2025 Feb 26;10(4):370-8. doi: 10.1001/jamacardio.2025.0016. Online ahead of print. PMID 40009358
- [Derived] Butt JH, Jhund PS, Henderson AD, Claggett BL, Desai AS, Viswanathan P, Kolkhof P, Schloemer P, Amarante F, Lam CSP, Senni M, Shah SJ, Voors AA, Zannad F, Pitt B, Vaduganathan M, Solomon SD, McMurray JJV; FINEARTS-HF Committees and Investigators. Finerenone and new-onset diabetes in heart failure: a prespecified analysis of the FINEARTS-HF trial. Lancet Diabetes Endocrinol. 2025 Feb;13(2):107-118. doi: 10.1016/S2213-8587(24)00309-7. Epub 2025 Jan 13. PMID 39818225
- [Derived] Butt JH, Henderson AD, Jhund PS, Claggett BL, Desai AS, Lay-Flurrie J, Viswanathan P, Lage A, Scheerer MF, Lam CSP, Senni M, Shah SJ, Voors AA, Bauersachs J, Fonseca C, Kosiborod MN, Linssen GCM, Petrie MC, Schou M, Verma S, Zannad F, Pitt B, Vaduganathan M, Solomon SD, McMurray JJV. Finerenone, Obesity, and Heart Failure With Mildly Reduced/Preserved Ejection Fraction: Prespecified Analysis of FINEARTS-HF. J Am Coll Cardiol. 2025 Jan 21;85(2):140-155. doi: 10.1016/j.jacc.2024.10.111. Epub 2024 Dec 10. PMID 39665701
- [Derived] Chimura M, Wang X, Jhund PS, Henderson AD, Claggett BL, Desai AS, Fonseca C, Goncalvesova E, Katova T, Mueller K, Glasauer A, Rohwedder K, Viswanathan P, Nodari S, Lam CSP, Saldarriaga CI, Senni M, Sharma K, Voors AA, Zannad F, Pitt B, Vardeny O, Vaduganathan M, Solomon SD, McMurray JJV. Finerenone in Women and Men With Heart Failure With Mildly Reduced or Preserved Ejection Fraction: A Secondary Analysis of the FINEARTS-HF Randomized Clinical Trial. JAMA Cardiol. 2025 Jan 1;10(1):59-70. doi: 10.1001/jamacardio.2024.4613. PMID 39550721
- [Derived] Vardeny O, Vaduganathan M, Claggett BL, Desai AS, Jhund PS, Lam CSP, Senni M, Shah SJ, Voors AA, Zannad F, Pitt B, Matsumoto S, Merkely B, Zieroth S, Yilmaz MB, Lay-Flurrie J, Viswanathan P, Horvat-Broecker A, Scalise A, McMurray JJV, Solomon SD. Finerenone, Serum Potassium, and Clinical Outcomes in Heart Failure With Mildly Reduced or Preserved Ejection Fraction. JAMA Cardiol. 2025 Jan 1;10(1):42-48. doi: 10.1001/jamacardio.2024.4539. PMID 39550716
- [Derived] Mc Causland FR, Vaduganathan M, Claggett BL, Kulac IJ, Desai AS, Jhund PS, Henderson AD, Brinker M, Perkins R, Scheerer MF, Schloemer P, Lam CSP, Senni M, Shah SJ, Voors AA, Zannad F, Pitt B, McMurray JJV, Solomon SD. Finerenone and Kidney Outcomes in Patients With Heart Failure: The FINEARTS-HF Trial. J Am Coll Cardiol. 2025 Jan 21;85(2):159-168. doi: 10.1016/j.jacc.2024.10.091. Epub 2024 Oct 25. PMID 39490700
- [Derived] Docherty KF, Henderson AD, Jhund PS, Claggett BL, Desai AS, Mueller K, Viswanathan P, Scalise A, Lam CSP, Senni M, Shah SJ, Voors AA, Zannad F, Pitt B, Vaduganathan M, Solomon SD, McMurray JJV. Efficacy and Safety of Finerenone Across the Ejection Fraction Spectrum in Heart Failure With Mildly Reduced or Preserved Ejection Fraction: A Prespecified Analysis of the FINEARTS-HF Trial. Circulation. 2025 Jan 7;151(1):45-58. doi: 10.1161/CIRCULATIONAHA.124.072011. Epub 2024 Sep 29. PMID 39342512
- [Derived] Vaduganathan M, Claggett BL, Kulac IJ, Miao ZM, Desai AS, Jhund PS, Henderson AD, Brinker M, Lay-Flurrie J, Viswanathan P, Scheerer MF, Lage A, Lam CSP, Senni M, Shah SJ, Voors AA, Zannad F, Pitt B, McMurray JJV, Solomon SD. Effects of the Nonsteroidal MRA Finerenone With and Without Concomitant SGLT2 Inhibitor Use in Heart Failure. Circulation. 2025 Jan 14;151(2):149-158. doi: 10.1161/CIRCULATIONAHA.124.072055. Epub 2024 Sep 28. PMID 39340828
- [Derived] Vaduganathan M, Claggett BL, Desai AS, Jhund PS, Lam CSP, Senni M, Shah SJ, Voors AA, Zannad F, Pitt B, Borentian M, Lay-Flurrie J, Viswanathan P, Behmenburg FU, McMurray JJV, Solomon SD. Estimated Long-Term Benefits of Finerenone in Heart Failure: A Prespecified Secondary Analysis of the FINEARTS-HF Randomized Clinical Trial. JAMA Cardiol. 2025 Feb 1;10(2):176-181. doi: 10.1001/jamacardio.2024.3782. PMID 39332395
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards — https://clinicaltrials.bayer.com/study/20103

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at multiple centers in 37 countries/regions between 14-Sep-2020 (first participant first visit) and 14-Jun-2024 (last participant last visit).
Pre-assignment Details: Of the 7463 screened participants, 1447 were screening failures, 6016 were randomized. Of the 3011 participants randomized into the finerenone group and the 3005 into the placebo group, 8 and 7 participants respectively were prospectively excluded from analysis due to major Good Clinical Practice (GCP) violations.
Groups:
- Finerenone (BAY94-8862): Participants received finerenone 10 mg, 20 mg or 40 mg once daily.
- Placebo: Participants received matching placebo once daily.
Period: Overall Study
Arm/Group | Finerenone (BAY94-8862) | Placebo
Started (randomized) | 3011 | 3005
Valid for FAS (valid for FAS (full analysis set)) | 3003 | 2998
Completed | 2996 | 2986
Not Completed | 15 | 19
Not completed — Lost to Follow-up | 1 | 5
Not completed — Withdrawal by Subject | 6 | 7
Not completed — major GCP violations | 8 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Finerenone (BAY94-8862) | Placebo | Total
Number analyzed (Participants) | 3003 | 2998 | 6001
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.94 (9.60) | 72.04 (9.69) | 71.99 (9.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1355 | 1377 | 2732
  Male | 1648 | 1621 | 3269
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 75 | 74 | 149
  Asian | 497 | 499 | 996
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 49 | 39 | 88
  White | 2366 | 2369 | 4735
  More than one race | 7 | 8 | 15
  Unknown or Not Reported | 8 | 9 | 17
NYHA class [Count of Participants; unit: Participants] — The New York Heart Association (NYHA) Functional Classification is a simple scale that classifies patients with heart failure based on the severity of their symptoms and how those symptoms affect their physical activity, which ranges from Class I to Class IV, a lower class number is indicative of a better condition.
  Participants
    NYHA class II | 2081 | 2065 | 4146
    NYHA class III | 903 | 910 | 1813
    NYHA class IV | 18 | 23 | 41
    missing | 1 | 0 | 1
Baseline LVEF [Mean (Standard Deviation); unit: percentage of ejection fraction] — LVEF: Left ventricular ejection fraction, which is used to assess how well the left ventricle of the heart pumps blood with each beat. A normal LVEF ranges from 55% to 70%. When the LVEF is below 55%, it suggests that the heart's pumping ability is reduced.
  percentage of ejection fraction | 52.64 (7.82) | 52.49 (7.81) | 52.56 (7.81)

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of the Composite Endpoint of Cardiovascular Death and Total (First and Recurrent) Heart Failure Events
Description: Number of composite endpoint events of cardiovascular death and total (first and recurrent) heart failure (HF) events (hospitalization for heart failure or urgent HF visit) in HF patients.
Time Frame: From randomization up until the end of study, with an average study duration of 32 months
Population: Full analysis set
Measure: Number; unit: events
Arm/Group | Finerenone (BAY94-8862) | Placebo
Number analyzed (Participants) | 3003 | 2998
events | 1083 | 1283
Statistical Analysis 1: Comparison: Finerenone (BAY94-8862) vs Placebo; Rate Ratio (Finerenone/Placebo); Test type: Superiority; p = 0.0072, stratified Andersen-Gill model — Two-sided p-value; p-value threshold =0.04967;; stratified Andersen-Gill model with robust sandwich estimate for the covariance matrix of recurrent events; Rate ratio = 0.84, 95% CI 2-sided [0.74 to 0.95] — stratified Andersen-Gill model with robust sandwich estimate for the covariance matrix of recurrent events

2. Primary Outcome: Occurrence of the Composite Endpoint of Cardiovascular Death and Total (First and Recurrent) Heart Failure Events
Description: Number of participants with composite endpoint events of cardiovascular death and total (first and recurrent) heart failure (HF) events (hospitalization for heart failure or urgent HF visit) in HF patients.
Time Frame: From randomization up until the end of study, with an average study duration of 32 months
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Finerenone (BAY94-8862) | Placebo
Number analyzed (Participants) | 3003 | 2998
Participants | 624 | 719

3. Secondary Outcome: Occurrence of Total (First and Recurrent) Heart Failure Events
Description: Number of total (first and recurrent) heart failure events.
Time Frame: From randomization up until the end of study, with an average study duration of 32 months
Population: Full analysis set
Measure: Number; unit: events
Arm/Group | Finerenone (BAY94-8862) | Placebo
Number analyzed (Participants) | 3003 | 2998
events | 842 | 1024
Statistical Analysis 1: Comparison: Finerenone (BAY94-8862) vs Placebo; Rate Ratio (Finerenone/Placebo); Test type: Superiority; p = 0.0062, Stratified Andersen-Gill model — Two-sided p-value; p-value threshold=0.04967;; stratified Andersen-Gill model with robust sandwich estimate for the covariance matrix of recurrent events; Rate ratio = 0.82, 95% CI 2-sided [0.71 to 0.94] — stratified Andersen-Gill model with robust sandwich estimate for the covariance matrix of recurrent events

4. Secondary Outcome: Occurrence of Total (First and Recurrent) Heart Failure Events
Description: Number of participants with total (first and recurrent) heart failure events.
Time Frame: From randomization up until the end of study, with an average study duration of 32 months
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Finerenone (BAY94-8862) | Placebo
Number analyzed (Participants) | 3003 | 2998
Participants | 479 | 573

5. Secondary Outcome: Change From Baseline in Total Symptom Score (TSS) of the Kansas City Cardiomyopathy Questionnaire (KCCQ)
Description: The Kansas City Cardiomyopathy Questionnaire Total Symptom Score (KCCQ-TSS) is ranged from 0 to 100. A higher score (closer to 100) reflects fewer symptoms, indicating better heart failure symptom status.
  For the change from baseline the combined and averaged result across the entire time frame is reported.
Time Frame: From baseline to Month 6, 9 and 12
Population: Full analysis set with available KCCQ measurements
Measure: Least Squares Mean (95% Confidence Interval); unit: score on scale
Arm/Group | Finerenone (BAY94-8862) | Placebo
Number analyzed (Participants) | 2731 | 2710
score on scale | 7.99 [7.37 to 8.62] | 6.43 [5.79 to 7.07]
Statistical Analysis 1: Comparison: Finerenone (BAY94-8862) vs Placebo; Difference in LS Mean; Test type: Other — mixed-effects model for repeated measures (MMRM); p < .0001, Mixed Models Analysis — Two-sided p-value;; The analysis was performed using mixed-effects model for repeated measures (MMRM); Difference in LS Mean = 1.56, 95% CI 2-sided [0.79 to 2.34]

6. Secondary Outcome: Proportion of Participants Who Showed Improvement in NHYA Class
Description: The New York Heart Association (NYHA) Functional Classification is a simple scale that classifies patients with heart failure based on the severity of their symptoms and how those symptoms affect their physical activity, which ranges from Class I to Class IV, a lower class number is indicative of a better condition. A patient was considered as having improved in NYHA class, if the NYHA class at Month 12 is at least one category improved compared to the baseline visit.
Time Frame: from baseline to Month 12
Population: Full analysis set with available NYHA measurement at baseline
Measure: Number (95% Confidence Interval); unit: Estimated proportion
Arm/Group | Finerenone (BAY94-8862) | Placebo
Number analyzed (Participants) | 3003 | 2998
Estimated proportion | 0.179 [0.163 to 0.195] | 0.178 [0.162 to 0.194]
Statistical Analysis 1: Comparison: Finerenone (BAY94-8862) vs Placebo; Odds ratio (finerenone /placebo); Test type: Other — Logistic regression analysis; p = 0.9295, Regression, Logistic — Two-sided p-value; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.88 to 1.15]

7. Secondary Outcome: First Occurrence of Renal Composite Events
Description: Number of participants with renal composite events encompassing the components sustained decrease in eGFR ≥50% relative to baseline over at least 4 weeks, sustained eGFR decline to <15 mL/min/1.73 m2 over at least 4 weeks, initiation of chronic dialysis and renal transplantation.
Time Frame: From randomization up to end of study visit, with an average study duration of 32 months
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Finerenone (BAY94-8862) | Placebo
Number analyzed (Participants) | 3003 | 2998
Participants | 75 | 55
Statistical Analysis 1: Comparison: Finerenone (BAY94-8862) vs Placebo; Cause-specific Hazard Ratio; Test type: Other — Stratified log-rank test; p = 0.1071, Stratified log-rank test — two-sided p-value; Cause-specific Hazard Ratio = 1.33, 95% CI 2-sided [0.94 to 1.89] — stratified Cox proportional hazards model

8. Secondary Outcome: Occurence of All-cause Mortality (Full Analysis Set)
Description: Number of participants with death due to any cause were reported as descriptive result. Number of participants with outcome death reported here includes deaths occurred after randomization until the end of the study visit. Deaths after end of study visit are not included in this table.
Time Frame: From randomization until end of study, with an average of 32 months
Population: Full analysis set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Finerenone (BAY94-8862) | Placebo
Number analyzed (Participants) | 3003 | 2998
Participants | 491 | 522
Statistical Analysis 1: Comparison: Finerenone (BAY94-8862) vs Placebo; Hazard Ratio; Test type: Other — Stratified log-rank test; p = 0.2794, stratified log-rank — two-sided p-value; cause-specific hazard ratio = 0.93, 95% CI 2-sided [0.83 to 1.06] — stratified Cox proportional hazards model

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events (TEAEs) are considered from the start of study intervention up to 3 days after the last study intervention administration, with an average treatment duration of 28 months. In contrast, numbers for all-cause mortality listed below consider all deaths after randomization over the entire average study duration of 32 months, independent of treatment and including deaths which occurred after the end of study visit in the 4-week follow-up period.
Description: The safety analysis set (SAF) included FAS participants who took ≥1 dose of study drug. 10 finerenone (n=3003) and 5 placebo participants (n=2998) took no drug, leaving 2993 in each SAF group. Heart failure and renal events were not counted as adverse events. All-cause mortality for FAS includes deaths from randomization to study end.
Groups:
- Placebo: Participants randomized to this group received matching placebo once daily.
- Never Received Treatment: Participants were randomized to either Finerenone or Placebo but never received study intervention.
Arm/Group | Finerenone (BAY94-8862) | Placebo | Never Received Treatment
All-Cause Mortality (participants affected / at risk) | 494/2993 | 528/2993 | 3/15
Serious Adverse Events (participants affected / at risk) | 1157/2993 | 1213/2993 | 0/15
Other Adverse Events (participants affected / at risk) | 1317/2993 | 1228/2993 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Finerenone (BAY94-8862) (N=2993) | Placebo (N=2993) | Never Received Treatment (N=15)
Anaemia (Blood and lymphatic system disorders) | 34 (42) | 31 (36) | 0 (0)
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 5 (5) | 6 (7) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Splenic haematoma (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Spontaneous haematoma (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Blood loss anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 0 (0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0)
Angina pectoris (Cardiac disorders) | 17 (23) | 26 (30) | 0 (0)
Angina unstable (Cardiac disorders) | 38 (43) | 36 (38) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 4 (4) | 5 (6) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 77 (95) | 73 (101) | 0 (0)
Atrial flutter (Cardiac disorders) | 14 (14) | 10 (10) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 6 (6) | 5 (5) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 5 (5) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 7 (7) | 9 (10) | 0 (0)
Cardiac amyloidosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac aneurysm (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 12 (12) | 11 (12) | 0 (0)
Cardiac failure (Cardiac disorders) | 18 (18) | 18 (20) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 5 (5) | 6 (6) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 4 (4) | 4 (4) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Conduction disorder (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cor pulmonale (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 20 (23) | 17 (17) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 6 (7) | 8 (8) | 0 (0)
Myocardial fibrosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 7 (7) | 9 (10) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0)
Pericardial effusion (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 3 (3) | 3 (3) | 0 (0)
Pericarditis constrictive (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0)
Sinoatrial block (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 4 (5) | 3 (6) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0)
Tachycardia paroxysmal (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 1 (3) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 4 (7) | 2 (3) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 2 (2) | 3 (3) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 8 (9) | 13 (18) | 0 (0)
Atrial thrombosis (Cardiac disorders) | 3 (4) | 0 (0) | 0 (0)
Cardiac pseudoaneurysm (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Bradyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiovascular deconditioning (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 2 (2) | 7 (7) | 0 (0)
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Dilated cardiomyopathy (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Tricuspid valve disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac valve disease (Cardiac disorders) | 1 (1) | 3 (4) | 0 (0)
Mitral valve disease (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Ventricular tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiorenal syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Microvascular coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 12 (13) | 10 (10) | 0 (0)
Chronic coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Dermoid cyst (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Familial amyloidosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Janus kinase 2 mutation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 5 (5) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Cushing's syndrome (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 8 (10) | 6 (6) | 0 (0)
Cataract subcapsular (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic eye disease (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 1 (2) | 0 (0)
Macular degeneration (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Open angle glaucoma (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Ophthalmoplegia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 3 (4) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Age-related macular degeneration (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Neovascular age-related macular degeneration (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal adhesions (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 6 (7) | 10 (10) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Acute abdomen (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (3) | 5 (5) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 6 (8) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (3) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 2 (3) | 1 (1) | 0 (0)
Gastrointestinal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 17 (17) | 8 (10) | 0 (0)
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 3 (3) | 5 (5) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 7 (8) | 14 (15) | 0 (0)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 5 (5) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 6 (6) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Obturator hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophageal achalasia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatic haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2) | 7 (7) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Proctitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 5 (5) | 3 (4) | 0 (0)
Rectal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 4 (5) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 (5) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 3 (3) | 0 (0)
Pancreatic mass (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 8 (9) | 3 (3) | 0 (0)
Enterocutaneous fistula (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 6 (6) | 3 (3) | 0 (0)
Acquired oesophageal web (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Salivary gland mass (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hernial eventration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Duodenogastric reflux (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Erosive duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal sphincter insufficiency (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Bile acid malabsorption (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestinal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal incarcerated hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Strangulated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Asthenia (General disorders) | 6 (6) | 4 (4) | 0 (0)
Chest discomfort (General disorders) | 2 (2) | 1 (1) | 0 (0)
Chest pain (General disorders) | 23 (31) | 22 (23) | 0 (0)
Condition aggravated (General disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 29 (29) | 52 (52) | 0 (0)
Fatigue (General disorders) | 2 (2) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 1 (1) | 0 (0)
Hernia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperpyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 1 (1) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 1 (1) | 0 (0)
Incarcerated hernia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 8 (8) | 0 (0)
Sudden death (General disorders) | 16 (16) | 17 (17) | 0 (0)
Sudden cardiac death (General disorders) | 14 (14) | 16 (16) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pacemaker generated arrhythmia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Polyp (General disorders) | 1 (1) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 3 (3) | 2 (2) | 0 (0)
Prosthetic cardiac valve thrombosis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Accidental death (General disorders) | 1 (1) | 1 (1) | 0 (0)
Medical device site haematoma (General disorders) | 0 (0) | 1 (1) | 0 (0)
Vascular stent stenosis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 4 (4) | 5 (5) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Alcoholic liver disease (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 2 (2) | 1 (1) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 2 (2) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 3 (3) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 4 (5) | 8 (8) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 7 (7) | 9 (10) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 5 (5) | 5 (5) | 0 (0)
Cirrhosis alcoholic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 3 (3) | 3 (4) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatitis alcoholic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Biliary dyskinesia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hydrocholecystis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic lesion (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Congestive hepatopathy (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Amyloidosis (Immune system disorders) | 3 (3) | 0 (0) | 0 (0)
Anaphylactic shock (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Anaphylactoid reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Primary amyloidosis (Immune system disorders) | 1 (1) | 1 (1) | 0 (0)
Sarcoidosis (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 6 (6) | 5 (5) | 0 (0)
Bacteraemia (Infections and infestations) | 4 (4) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 13 (14) | 11 (15) | 0 (0)
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 17 (18) | 24 (25) | 0 (0)
Dacryocystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 4 (4) | 0 (0)
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Encephalomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Endocarditis staphylococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Epididymitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 4 (4) | 4 (6) | 0 (0)
Escherichia sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Fournier's gangrene (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 2 (2) | 6 (6) | 0 (0)
Gas gangrene (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 6 (6) | 6 (6) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Infected skin ulcer (Infections and infestations) | 2 (3) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 7 (7) | 5 (5) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 6 (6) | 7 (8) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 3 (3) | 4 (4) | 0 (0)
Osteomyelitis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis chronic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 2 (2) | 3 (3) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 87 (98) | 110 (116) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 2 (2) | 5 (5) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia legionella (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Pneumonia moraxella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 2 (2) | 5 (5) | 0 (0)
Postoperative wound infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Prostatic abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Pyoderma (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyonephrosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Salmonellosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 25 (25) | 16 (16) | 0 (0)
Septic arthritis staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 7 (7) | 9 (9) | 0 (0)
Skin infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Subacute endocarditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Tuberculosis of intrathoracic lymph nodes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tuberculous pleurisy (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 4 (4) | 0 (0)
Urinary tract infection (Infections and infestations) | 29 (31) | 26 (28) | 0 (0)
Urinary tract infection enterococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 3 (3) | 2 (2) | 0 (0)
Urosepsis (Infections and infestations) | 5 (5) | 5 (5) | 0 (0)
Bursitis infective staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 3 (3) | 2 (2) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 6 (6) | 0 (0)
Coronavirus infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Candida pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Citrobacter sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Subdiaphragmatic abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Emphysematous cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Psoas abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 5 (5) | 0 (0)
Infective tenosynovitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Biliary sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Abdominal sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Intervertebral discitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Diabetic foot infection (Infections and infestations) | 3 (3) | 2 (2) | 0 (0)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 7 (8) | 6 (6) | 0 (0)
Clostridial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Escherichia infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 8 (8) | 10 (10) | 0 (0)
Cholecystitis infective (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Infective spondylitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Acarodermatitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tongue abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rotavirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Streptococcal endocarditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Meningoencephalitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Medical device site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Medical device site joint infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Systemic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pulmonary paracoccidioidomycosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Vascular device infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
H3N2 influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Large intestine infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Infected gouty tophus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 69 (69) | 71 (73) | 0 (0)
Diverticulitis intestinal perforated (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 28 (28) | 30 (30) | 0 (0)
Suspected COVID-19 (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
SARS-CoV-2 sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Norovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Klebsiella urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Accident (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Extradural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 15 (15) | 14 (14) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 4 (4) | 9 (9) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 15 (15) | 17 (17) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 4 (4) | 0 (0)
Heat stroke (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 12 (12) | 7 (7) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 9 (9) | 0 (0)
Hyphaema (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (2) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 4 (5) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0)
Pulmonary contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 5 (5) | 8 (8) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Snake bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 6 (6) | 4 (4) | 0 (0)
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 4 (5) | 2 (2) | 0 (0)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 8 (9) | 9 (9) | 0 (0)
Synovial rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0)
Shoulder fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 6 (6) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 3 (3) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 0 (0)
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Shunt stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Incision site haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Postpericardiotomy syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 7 (7) | 6 (6) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (3) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0)
Shunt aneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 4 (4) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal column injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 5 (5) | 4 (4) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Adjacent segment degeneration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Craniofacial fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Nasal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Injury of conjunctiva (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Biopsy prostate (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase MB increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Carcinoembryonic antigen increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Heart rate decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Intraocular pressure decreased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Ureteroscopy (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Weight increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 3 (3) | 0 (0)
Anticoagulation drug level above therapeutic (Investigations) | 1 (1) | 0 (0) | 0 (0)
Renal function test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Occult blood positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
Angiocardiogram (Investigations) | 2 (2) | 1 (1) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 2 (2) | 2 (2) | 0 (0)
Computerised tomogram heart abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Alkalosis hypochloraemic (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 14 (16) | 6 (8) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 3 (3) | 3 (3) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 3 (3) | 8 (10) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 19 (19) | 6 (7) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 9 (11) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 10 (11) | 3 (5) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Marasmus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0)
Mineral metabolism disorder (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 4 (4) | 3 (3) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 0 (0)
Adult failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 7 (7) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (10) | 8 (8) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (6) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (4) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 9 (9) | 11 (13) | 0 (0)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Scleroderma (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Neck mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (6) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Connective tissue inflammation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Connective tissue disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Immobilisation syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (5) | 0 (0)
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
B-cell small lymphocytic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3) | 0 (0)
Benign neoplasm of adrenal gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 6 (6) | 0 (0)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Carcinoma in situ of penis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 6 (6) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3) | 0 (0)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (3) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Mediastinum neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (5) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0)
Papillary serous endometrial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Sarcoma uterus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastases to salivary gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Retroperitoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 10 (12) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (11) | 9 (9) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Malignant mediastinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Paraganglion neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Lip neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung infiltration malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Rosai-Dorfman syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Ovarian cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Laryngeal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (4) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 0 (0)
Ovarian granulosa cell tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Intraductal papillary-mucinous carcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Myeloproliferative neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Neuroendocrine tumour of the lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Follicular lymphoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Malignant gastric ulcer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Bell's palsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 4 (5) | 3 (5) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral artery occlusion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dementia (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 12 (12) | 7 (7) | 0 (0)
Drop attacks (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Epilepsy (Nervous system disorders) | 3 (4) | 0 (0) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertensive encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Intraventricular haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 2 (2) | 5 (5) | 0 (0)
Movement disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Myelopathy (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Parkinsonism (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0)
Quadriplegia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Radiculopathy (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0)
Sciatica (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 4 (4) | 1 (1) | 0 (0)
Spondylitic myelopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 2 (2) | 6 (6) | 0 (0)
Syncope (Nervous system disorders) | 25 (26) | 22 (23) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 8 (8) | 7 (7) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Wernicke's encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Quadriparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal epidural haematoma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular insufficiency (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Vascular encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Orthostatic intolerance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Brain injury (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Lumbosacral radiculopathy (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Post cardiac arrest syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Thoracic radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Alcoholic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 3 (3) | 1 (1) | 0 (0)
Conversion disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Disorientation (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Eating disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Mania (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 2 (2) | 2 (3) | 0 (0)
Suicidal behaviour (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Somatic symptom disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mixed anxiety and depressive disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Anuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 6 (6) | 5 (5) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Intercapillary glomerulosclerosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 2 (5) | 1 (2) | 0 (0)
Nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 8 (8) | 5 (5) | 0 (0)
Renal infarct (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 6 (7) | 3 (3) | 0 (0)
Urinary tract disorder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0)
Postrenal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 10 (10) | 11 (11) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 7 (7) | 6 (6) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 54 (56) | 28 (30) | 0 (0)
Prerenal failure (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0)
Subcapsular renal haematoma (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 6 (6) | 3 (3) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Scrotal swelling (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Ovarian haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 17 (18) | 0 (0)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 2 (3) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 18 (20) | 27 (32) | 0 (0)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 (17) | 13 (13) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 10 (10) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 8 (10) | 0 (0)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Malignant pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 (9) | 11 (13) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 12 (13) | 5 (5) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (6) | 0 (0)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 9 (10) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acquired diaphragmatic eventration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
Bronchial wall thickening (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Skin erosion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 4 (4) | 6 (9) | 0 (0)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (5) | 0 (0)
Immobile (Social circumstances) | 0 (0) | 1 (1) | 0 (0)
Angioplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Aortic valve replacement (Surgical and medical procedures) | 1 (1) | 2 (2) | 0 (0)
Appendicectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Bladder calculus removal (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Cardiac pacemaker insertion (Surgical and medical procedures) | 8 (8) | 4 (4) | 0 (0)
Cardiac pacemaker removal (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Cardioversion (Surgical and medical procedures) | 2 (2) | 3 (3) | 0 (0)
Carotid endarterectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0)
Cryotherapy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Glossectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 5 (5) | 2 (2) | 0 (0)
Inguinal hernia repair (Surgical and medical procedures) | 5 (5) | 0 (0) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 3 (4) | 2 (2) | 0 (0)
Leg amputation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Pelvic floor repair (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Renal stone removal (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Spinal laminectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Toe amputation (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0)
Transurethral prostatectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Umbilical hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Ureteric calculus removal (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0)
Urethrotomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Cardiac pacemaker replacement (Surgical and medical procedures) | 4 (4) | 4 (4) | 0 (0)
Implantable defibrillator insertion (Surgical and medical procedures) | 1 (2) | 1 (1) | 0 (0)
Knee operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Shoulder arthroplasty (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0)
Coronary angioplasty (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0)
Hip surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Coronary arterial stent insertion (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Cholelithotomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Polypectomy (Surgical and medical procedures) | 0 (0) | 2 (2) | 0 (0)
Rehabilitation therapy (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0)
Renal artery angioplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Peripheral artery angioplasty (Surgical and medical procedures) | 1 (2) | 1 (1) | 0 (0)
Peripheral nerve decompression (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Cardiac resynchronisation therapy (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0)
Cardiac ablation (Surgical and medical procedures) | 3 (3) | 2 (2) | 0 (0)
Haematoma evacuation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Cardiac operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Colectomy (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0)
Prostatectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Gastrectomy (Surgical and medical procedures) | 0 (0) | 2 (2) | 0 (0)
Retinal operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Shoulder operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Percutaneous coronary intervention (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0)
Intraocular lens implant (Surgical and medical procedures) | 1 (2) | 0 (0) | 0 (0)
Eventration repair (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Transcatheter aortic valve implantation (Surgical and medical procedures) | 0 (0) | 2 (2) | 0 (0)
Metabolic surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Atrial appendage closure (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Drug titration (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Accelerated hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 4 (4) | 2 (2) | 0 (0)
Aortic dissection (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 4 (4) | 7 (8) | 0 (0)
Arterial thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Blood pressure fluctuation (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Embolism arterial (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Essential hypertension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Femoral artery aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 2 (2) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 7 (8) | 11 (11) | 0 (0)
Hypertensive crisis (Vascular disorders) | 4 (4) | 7 (7) | 0 (0)
Hypotension (Vascular disorders) | 12 (14) | 9 (9) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 2 (2) | 1 (1) | 0 (0)
Intermittent claudication (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 4 (4) | 7 (7) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 5 (5) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 2 (3) | 0 (0)
Thrombosis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Varicose ulceration (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Labile hypertension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 2 (2) | 0 (0)
Dry gangrene (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 2 (2) | 0 (0)
Hypertensive emergency (Vascular disorders) | 3 (3) | 4 (4) | 0 (0)
Hypertensive urgency (Vascular disorders) | 0 (0) | 3 (3) | 0 (0)
Extremity necrosis (Vascular disorders) | 0 (0) | 2 (4) | 0 (0)
Arterial haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic vascular disorder (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 10 (13) | 8 (12) | 0 (0)
Aortic arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Aortic dissection rupture (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Subgaleal haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Obstructive shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral venous disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Brachiocephalic arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Brachiocephalic artery stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Device malfunction (Product Issues) | 3 (3) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 3 (3) | 0 (0) | 0 (0)
Device fastener issue (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Device inappropriate shock delivery (Product Issues) | 1 (1) | 1 (1) | 0 (0)
Device loosening (Product Issues) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Finerenone (BAY94-8862) (N=2993) | Placebo (N=2993) | Never Received Treatment (N=15)
Anaemia (Blood and lymphatic system disorders) | 169 (193) | 162 (178) | 0 (0)
Cardiac failure (Cardiac disorders) | 116 (143) | 168 (218) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 167 (208) | 129 (157) | 0 (0)
Urinary tract infection (Infections and infestations) | 150 (184) | 149 (194) | 0 (0)
COVID-19 (Infections and infestations) | 292 (301) | 297 (318) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 156 (219) | 107 (144) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 252 (348) | 107 (139) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 88 (105) | 196 (255) | 0 (0)
Dizziness (Nervous system disorders) | 170 (198) | 137 (158) | 0 (0)
Renal impairment (Renal and urinary disorders) | 193 (232) | 110 (127) | 0 (0)
Hypertension (Vascular disorders) | 103 (121) | 179 (215) | 0 (0)
Hypotension (Vascular disorders) | 210 (240) | 128 (143) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-05-16): https://cdn.clinicaltrials.gov/large-docs/26/NCT04435626/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-20): https://cdn.clinicaltrials.gov/large-docs/26/NCT04435626/SAP_001.pdf